

# STATISTICAL ANALYSIS PLAN

An Open-Label, Phase 1b/2 Study to Evaluate the Safety and Efficacy of Fruquintinib in Combination with Tislelizumab in Patients with Advanced Solid Tumors

Protocol Number: 2020-013-00US3

Name of Test Drug: Fruquintinib (HMPL-013)

Tislelizumab (BGB-A317)

Phase: Phase 1b/2

Sponsor Name: HUTCHMED Limited

Building 4, 720 Cailun Road, China (Shanghai) Pilot Free Trade Zone

Shanghai, China, 201203

Phone: PPD

http://www.hutch-med.com

Analysis Plan Version Version 2.0

Effective Date 29 July 2024

**Compliance:** The study described in this report was performed according to the principle of Good Clinical Practice (GCP).

#### Confidentiality Statement

The information contained in this document is the confidential and proprietary information of HUTCHMED Limited and its affiliates and except as may be required by applicable laws or regulation, may not be disclosed to others without prior written permission of HUTCHMED Limited.

# APPROVAL SIGNATURES

# AUTHOR:

APPROVED BY:



# REVISION HISTORY

| Date | Version | Description | Author |
|---|---|---|---|
| 10Jun2021 | 0.1 | Initial version | PPD |
| 01July2021 | 0.2 | Updated due to SR and internal Syneos | PPD |
| | | review. Version sent to HMP | |
| 18Oct2021 | 0.3 | Updated due to HMP comments and | PPD |
| | | protocol amendment 2 | |
| 15Dec2021 | 0.4 | Updated due to HMP comments | PPD |
| 04Mar2022 | 0.5 | Updated due to HMP comments and | PPD |
| | | protocol amendment 3 | |
| 28Mar2022 | 1.0 | Updated due to HMP comments and finalized | PPD |
| 21Jul2022 | 1.1 | Update sponsor name to HUTCHMED Limited and the relevant address information Updated MedDRA dictionary version and | |
| | | WHO Drug dictionary version. | |
| | | Added some additional hepatic criteria<br>in section 4.4.3 | |
| | | Updated visit windowing table 11 in section 5.1.3. | |
| | | Removed in section 5.2.1 the derivation of EOS reasons as it is now reported in the CRF. | |
| | | Updated section 5.4.1 (Pharmacokinetic analysis) and 5.4.2 (Immunogenicity analysis). | |
| | | Updated Appendix 1: Study<br>Schedule of Events | |
| | | Updated Appendix 5: Updated<br>MedDRA Preferred Term List using<br>version 25.0 | |
| | | Added Appendix 6 to define COVID related AEs | |

| | | Added Appendix 7 to define conversion | |
|---|---|---|---|
| | | tables for urinalysis results | |
| 29Jul2024 | 2.0 | Update due to HMP comments and protocol amendment 4 dated 02 February 2023 and amendment 5 dated 06 December 2023. Update prior to the Database Lock. - Updated the DLT-Evaluable Analysis Set and PK Analysis Set definitions Removed Appendix 5 Considerations for assigning response category and patients without any post-baseline tumor assessment (patients who died or | PPD |
| | | progressed clinically prior to the first scheduled tumor assessment) were added in Sections 4.2.1 and 4.2.2. Details on censoring for PFS were added in Table 3. Text in Section 6.2 was aligned with the interim analyses performed during the study conduct. Additional details provided on | |
| | | presentation of PK data in<br>Section 4.5.1 and ADA data in<br>Section 4.5.2. | |

# TABLE OF CONTENTS

| TABLE | JF CONTENTS | |
|----------|-----------------------------------------------------|----|
| LIST OF | TABLES | 8 |
| LIST OF | ABBREVIATIONS | 9 |
| 1. | INTRODUCTION | 11 |
| 2. | STUDY DETAILS | 12 |
| 2.1. | Study Objectives | 12 |
| 2.2. | Study Design | 14 |
| 2.3. | Determination of Sample Size | 17 |
| 3. | ANALYSIS SETS | 19 |
| 3.1. | Definition of Analysis Sets | 19 |
| 3.1.1. | Enrolled Set | 19 |
| 3.1.2. | Safety Analysis Set | 19 |
| 3.1.3. | DLT-Evaluable Analysis Set | 19 |
| 3.1.4. | Response Evaluable Analysis Set | 19 |
| 3.1.5. | Pharmacokinetics (PK) Analysis Set | 19 |
| 3.1.6. | Antidrug Antibody (ADA) Analysis Set | 19 |
| 3.2. | Protocol Deviation | 19 |
| 4. | ENDPOINTS | 20 |
| 4.1. | General Principles for Derived and Transformed Data | 20 |
| 4.1.1. | Reference Start Date and End Date and Study Day | 20 |
| 4.1.2. | Baseline and Change from Baseline | 20 |
| 4.1.3. | Treatment Period | 20 |
| 4.2. | Efficacy Endpoints | 21 |
| 4.2.1. | Primary Endpoint | 21 |
| 4.2.2. | Secondary Endpoints | 22 |
| 4.2.2.1. | Progression-free Survival (PFS) | 22 |
| 4.2.2.2. | Disease Control Rate | 23 |
| 4.2.2.3. | Clinical Benefit Rate | 24 |

Date: 29 July 2024

| 4.2.2.4. | Duration of Response | 24 |
|----------|--------------------------------------------------------------|----|
| 4.2.2.5. | Overall Survival | 24 |
| 4.3. | Exposure Endpoints | 25 |
| 4.4. | Safety Endpoints | 27 |
| 4.4.1. | Dose Limiting Toxicities (DLTs) or DLT-equivalent | 27 |
| 4.4.2. | Adverse Events (AEs) | 27 |
| 4.4.3. | Laboratory | 29 |
| 4.4.4. | ECG | 31 |
| 4.4.5. | Vital Signs | 32 |
| 4.4.6. | Performance Status | 32 |
| 4.4.7. | Echocardiogram | 33 |
| 4.4.8. | Physical Examination | 33 |
| 4.5. | Other Endpoints | 33 |
| 4.5.1. | Pharmacokinetic Endpoint | 33 |
| 4.5.2. | Immunogenicity | 33 |
| 4.5.3. | Exploratory Endpoints | 33 |
| 5. | ANALYSIS METHODS | 34 |
| 5.1. | General Principles | 34 |
| 5.1.1. | General Methodology | 34 |
| 5.1.2. | Handling Missing Data | 35 |
| 5.1.2.1. | Adverse Events Start/End Date | 35 |
| 5.1.2.2. | Concomitant Medication/Procedure/Surgery Start/End Date | 36 |
| 5.1.2.3. | Subsequent Anti-Cancer Therapy Date | 37 |
| 5.1.2.4. | Primary Diagnosis Date and Metastatic Disease Diagnosis Date | 37 |
| 5.1.3. | Visit Windowing | 37 |
| 5.1.4. | Adjustment of Covariates | 41 |
| 5.2. | Analysis Methods | 41 |
| 5.2.1. | Patient Disposition | 41 |
| 5.2.2. | Protocol Deviation | 41 |

| 5.2.3. | Demographic and Other Baseline Characteristics | 41 |
|-----------|-------------------------------------------------------|----|
| 5.2.4. | Disease Characteristics | 42 |
| 5.2.5. | Medical History | 42 |
| 5.2.6. | Prior and Subsequent Anti-Cancer Therapy | 42 |
| 5.2.6.1. | Prior and Subsequent Anti-Cancer Medication | 43 |
| 5.2.6.2. | Prior and Subsequent Anti-Cancer Radiotherapy | 43 |
| 5.2.6.3. | Prior and Subsequent Anti-Cancer Procedure or Surgery | 43 |
| 5.2.7. | Prior and Concomitant Medications | 44 |
| 5.2.8. | Concomitant Procedure | 44 |
| 5.2.9. | Efficacy Analyses | 44 |
| 5.2.9.1. | Primary Efficacy Analyses | 45 |
| 5.2.9.2. | Secondary Efficacy Analyses | 45 |
| 5.2.9.3. | Sensitivity Analysis for Efficacy Endpoint | 45 |
| 5.2.10. | Exposure of Study Treatment | 45 |
| 5.2.11. | Safety Analyses | 46 |
| 5.2.11.1. | Dose-Limiting Toxicity (DLT) | 46 |
| 5.2.11.2. | Adverse Events | 46 |
| 5.2.11.3. | Death | 48 |
| 5.2.11.4. | Laboratory Evaluations | 48 |
| 5.2.11.5. | ECG | 49 |
| 5.2.11.6. | Vital Signs | 49 |
| 5.2.11.7. | Performance Status | 49 |
| 5.2.11.8. | Echocardiogram | 49 |
| 5.2.11.9. | Physical Examination | 49 |
| 5.3. | Subgroup Analyses | 49 |
| 5.4. | Other Analyses | 49 |
| 5.4.1. | Pharmacokinetic Analysis | 49 |
| 5.4.1.1. | Handling of Missing Data | 50 |
| 5.4.1.2. | Handling of Dose Reduction or Interruption. | 50 |

| 5.4.1.3. | Handling of below the lower limit of quantification (BLQ) Data | 50 |
|---|---|---|
| 5.4.1.4. | Summary of PK concentration Data | 50 |
| 5.4.1.5. | Handling of the Difference between the Scheduled (nominal time) and the Actual Sampling Times (actual time) | 51 |
| 5.4.2. | Immunogenicity Analysis | 51 |
| 5.4.3. | Exploratory Analyses | 52 |
| 6. | PLANNED ANALYSIS | 53 |
| 6.1. | Independent Safety Data Monitoring | 53 |
| 6.2. | Interim Analysis | 53 |
| 6.3. | Final Analysis | 53 |
| 7. | CHANGE FROM THE PROTOCOL | 54 |
| REFERE | NCE | 55 |
| APPEND | IX | 56 |
| | List of Tables | |
| Table 1 | Estimated ORR and 2-Sided 95% Confidence Intervals | 18 |
| Table 2 | Best Overall Response When Confirmation of CR and PR are Required | 21 |
| Table 3 | Censoring Rules for PFS | 23 |
| Table 4 | Algorithms for Calculating Parameters Relevant to the Dose Exposure and Intensity | 26 |
| Table 5 | MedDRA Terms Used for Adverse Events of Special Interest | 28 |
| Table 6 | Laboratory Assessment | 29 |
| Table 7 | Potentially Clinically Significant Criteria for ECG. | 31 |
| Table 8 | Potentially Clinically Significant Criteria for Vital Signs | 32 |
| Table 10 | Treatment/Cohort Display in TLFs | 34 |
| Table 11 | Visit Windowing | 39 |

# LIST OF ABBREVIATIONS

| Abbreviation | Term |
|-----------------|------------------------------------------------|
| ADA | Antidrug Antibody |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ASCO | American Society for Clinical Oncology |
| ATC | Anatomic Therapeutic Classification |
| BLQ | Below the Lower Limit of Quantification |
| BMI | Body Mass Index |
| CAP | College of American Pathologists |
| CBR | Clinical Benefit Rate |
| CFB | Change from Baseline |
| CI | Confidence Interval |
| CR | Complete Response |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CYP3A | Cytochrome P450, family 3, subfamily A |
| DBL | Database Lock |
| DBP | Diastolic Blood Pressure |
| DCR | Disease Control Rate |
| DLT | Dose-limiting Toxicity |
| DoR | Duration of Response |
| DMC | Data Monitoring Committee |
| EC | Endometrial Cancer |
| ECG | Electrocardiogram |
| ECHO | Echocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| EOC | End of Cycle |
| EOI | End of Infusion |
| EOT | End of Treatment |
| ER/PR or ER/PGR | Estrogen Receptor/Progesterone Receptor |
| ICH | International Council on Harmonization |
| ICI | Immune Checkpoint Inhibitor |
| imAE | Immune-mediated AE |
| IO | Immuno-oncology |

| Abbreviation | Term |
|---|---|
| LLOQ | Lower Limit of Quantification |
| mCRC | Metastatic Colorectal Cancer |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MSI | Microsatellite Instability |
| MSS | Microsatellite Stable |
| NCI CTCAE | National Cancer Institute Common Terminology Criteria for Adverse |
| | Event |
| ORR | Objective Response Rate |
| OS | Overall Survival |
| PFS | Progression-free Survival |
| PD-L1 | Programmed Death Ligand 1 |
| PT | Preferred Term |
| RECIST 1.1 | Response Evaluation Criteria in Solid Tumors, Version 1.1 |
| RP2D | Recommended Phase 2 Dose |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| StdDev | Standard Deviation |
| SMQs | Standardized MedDRA Queries |
| SOC | System Organ Class |
| SRC | Safety Review Committee |
| TEAE | Treatment-emergent Adverse Event |
| TLF | Table, Listing, Figure |
| TNBC | Triple Negative Breast Cancer |
| TPR | Timepoint Response |
| WHO-DD | World Health Organization Drug Dictionary |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the planned statistical analyses and data presentations for study 2020-013-00US3. The SAP is based on the Protocol Amendment 5, dated 06 December 2023. Study measurements and assessments, planned statistical methods, and derived variables are summarized in this plan. Planned tables, figures, and listings are specified. All decisions regarding final analyses, as defined in this SAP document, have been made prior to locking the database. Any deviations from these guidelines will be documented in the clinical study report (CSR).

This is an amendment to the approved SAP (dated 21 July 2022) based on the most recent Protocol Amendment 5 dated 06 December 2023. Upon implementation of Protocol Amendment #4, enrollment to expansion cohorts A (TNBC immuno-oncology [IO]-treated in the metastatic setting), B (TNBC IO-Naïve in the metastatic setting) and C (EC IO Naïve) in this study has been permanently discontinued based upon the strategic evaluation of the clinical development of fruquintinib in the United States with HUTCHMED as the study Sponsor. For Cohort D (MSS mCRC, IO Naïve), at the time of this decision making, the enrollment was completed. This change is not based on any concern for patient safety or efficacy relative to fruquintinib and/or tislelizumab treatment. Patients who are currently enrolled in these cohorts and are deriving benefit from treatment with fruquintinib and/or tislelizumab may continue to participate in the study as per protocol. There is no planned interruption in the supply of fruquintinib or tislelizumab to clinical trial sites with active patients.

Syneos Health is to list and tabulate concentration data for fruquintinib, its metabolite M11, tislelizumab. Immunogenicity data will also be tabulated. Syneos Health are responsible for the production and quality control of all Study Data Tabulation Model (SDTM) datasets, Analysis Data Model (ADaM) datasets, and the tables, listings, and figures (TLFs) associated with these datasets. The SAP for population PK will be prepared in a separate analysis plan by another contract research organization (CRO).

# 2. STUDY DETAILS

# 2.1. Study Objectives

| Part | Tier | Objectives | Endpoints |
|---|---|---|---|
| Part 1:<br>Safety<br>Lead-in<br>Phase | Primary | To assess the safety and tolerability of fruquintinib in combination with tislelizumab in patients with advanced solid tumors | Adverse events (AEs) characterized by type, frequency, severity per The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0, timing, seriousness, relationship to study drug(s), and discontinuation of study drug(s) due to AEs |
| | | To confirm the recommended phase 2 dose (RP2D) of fruquintinib in combination with tislelizumab | RP2D |
| | Secondary | To evaluate the efficacy of fruquintinib<br>in combination with tislelizumab per<br>investigator assessment | objective response rate (ORR) progression free survival (PFS), disease control rate (DCR), clinical benefit rate (CBR), duration of response (DoR) overall survival (OS) |
| | | To characterize the PK profile of fruquintinib and metabolite M11 when combined with tislelizumab | Plasma concentrations of fruquintinib<br>and M11 |
| | | To evaluate the PK and immunogenicity of fruquintinib in combination with tislelizumab | Serum concentrations of tislelizumab<br>and incidence of anti-drug antibody<br>(ADA) to tislelizumab |
| Part 2:<br>Dose<br>Expansion<br>Phase | Primary | To evaluate the ORR assessed by the investigator in patients with advanced or metastatic TNBC, EC, or MSS mCRC when treated with fruquintinib in combination with tislelizumab | ORR per response evaluation criteria in solid tumors version 1.1 (RECIST v1.1) |
| | Secondary | To further evaluate efficacy of fruquintinib in combination with tislelizumab in patients with advanced or metastatic TNBC, EC, or MSS mCRC per investigator assessment | PFS, DCR, CBR, DoR, and OS |
| | | To characterize the safety of fruquintinib in combination with tislelizumab | AEs characterized by type, frequency, severity per NCI CTCAE v5.0, timing, seriousness, relationship to study drug(s), and discontinuation of study drug(s) due to AEs. |

| Part | Tier | Objectives | Endpoints |
|---|---|---|---|
| | | To assess the pharmacokinetic (PK) profile of fruquintinib and metabolite (M11) when combined with tislelizumab | Plasma concentrations and derived PK parameters of fruquintinib and M11. |
| | | To characterize the PK and immunogenicity of fruquintinib when combined with tislelizumab | Serum concentrations of tislelizumab<br>and incidence of ADA to tislelizumab |
| | | To detect the expression of programmed death-ligand (PD-L1), MSS/MSI status, and other biomarkers in tumor tissues of patients, and to perform relevant efficacy analysis to provide reference for the determination of dominant population | Changes from baseline in biomarkers<br>markers, correlation with drug exposure,<br>and association with efficacy and safety<br>parameters |
| | Exploratory | To explore potential biomarkers<br>associated with anti-tumor effects of<br>fruquintinib in combination with<br>tislelizumab | Changes from baseline in tumor markers,<br>correlation with drug exposure, and<br>association with efficacy and safety<br>parameters |

## 2.2. Study Design

This is an open-label, multicenter, non-randomized, phase 1b/2 study to assess the safety and efficacy of fruquintinib in combination with tislelizumab in patients with advanced or metastatic solid tumors. This study will be conducted in 2 parts: a Safety Lead-in phase (Part 1) and a dose expansion phase (Part 2). The overall study schematic is presented in Figure 1.

Figure 1 Study Design Schema



2L=second line; 3L=third line; EC=endometrial cancer; ECOG=Eastern Cooperative Oncology Group; IO=immune-oncology; mCRC=metastatic colorectal cancer; MSS=microsatellite stable; n=total number of patients; PS=performance status; QD=once daily; Q4W=every 4 weeks; RP2D=recommended Phase 2 dose; TNBC=triple negative breast cancer.

#### Part 1: Safety Lead-in Phase

Approximately 6 to 12 patients with histologically or cytologically documented advanced or metastatic solid tumors of any type who have progressed on standard systemic therapy and for which no effective therapy or standard of care exists will be enrolled and assessed for DLTs during the 28-day period DLT observation period. Patients may be either immuno-oncology (IO) treated or naïve in the metastatic setting. Patients with TNBC in the Safety Lead-in must meet eligibility criteria defined in cohorts A or B, and those with EC in the Safety Lead-in must meet eligibility criteria defined in cohort C.

Part 1 of the study will begin by enrolling the first 6 patients and evaluating for DLTs during the DLT observation period. Study drug administration will begin at the full dose of

fruquintinib (5 mg daily, 3 weeks on followed by 1 week off every 4-week cycle) in combination with tislelizumab (300 mg once every 4 weeks). A lower dose level of fruquintinib (4 mg daily, 3 weeks on followed by 1 week off every 4-week cycle) will be explored as necessary depending on observed toxicity.

Only dose limiting toxicities (DLTs) during the first cycle of treatment will be assessed.

- If 0 or 1 of 6 patients experiences a DLT, the study may proceed at the current dose
  of both drugs.
- If 2 or more patients experience a DLT, then, following consultation with the safety review committee (SRC), the study will proceed with enrollment in the next defined lower dose (Dose Level -1), an additional 6 patients will be enrolled, and the 28-day DLT observation period will be repeated.
- If 2 or more patients experience a DLT in Dose Level -1, enrollment in the study will cease.

### Part 2: Dose Expansion Phase

Approximately 140 patients will be enrolled, including approximately 60 patients with TNBC (approximately 30 patients in each cohort [A and B]) and approximately 40 patients with EC in Cohort C, and approximately 40 patients with MSS mCRC in Cohort D. Patients will be enrolled to one of the following 4 cohorts. Of note, based upon the strategic evaluation of the clinical development of fruquintinib, patient enrollment has been permanently discontinued for all cohorts in the dose expansion phase. At the time of deciding on discontinuation of enrollment, the Cohort D had completed the enrollment. Hence, the final actual total number of patients will reflect this strategic decision.

Cohort A (TNBC, immuno-oncology [IO]-treated in the metastatic setting):
 Patients must have histologically or cytologically documented, advanced or metastatic
 TNBC as defined by American Society for Clinical Oncology (ASCO)-College of
 American Pathologists (CAP) guidelines. Up to 15 patients in cohort A can have ER or
 PR low positive disease as defined by ASCO-CAP guidelines, if the treating physician
 considers the patient not eligible for adjuvant endocrine therapy. TNBC is defined as
 ER/PR positivity of <1%, and ER/PR low positive disease is defined by ER/PR positivity
 of 1% to 10% (Allison 2020).</p>

Patients must have progressed on at least 1 line, but no more than 3 lines, of cytotoxic therapy in the locally advanced or metastatic setting. Patients must have also progressed on prior immunotherapy in the metastatic setting (Rakha 2014)Rakha 2014.

Cohort B (TNBC, IO-Naïve in the metastatic setting):
 Patients must have histologically or cytologically documented, locally advanced or metastatic TNBC as defined by ASCO-CAP guidelines. Up to 15 patients in cohort B can have ER or PR low positive disease as defined by ASCO-CAP guidelines, if the treating physician considers the patient not eligible for adjuvant endocrine therapy.

TNBC is defined as ER/PR positivity of <1%, and ER/PR low positive disease is defined by ER/PR positivity of 1% to 10%.

Patients must have progressed on at least 1 line, but no more than 3 lines, of cytotoxic therapy in the locally advanced or metastatic setting. Patients must not have received prior therapy with an ICI or other immunotherapy in the metastatic setting.

### Cohort C (EC, IO Naïve):

Patients must have histologically or cytologically documented, advanced or metastatic EC.

Patients must have progressed on 1 prior, platinum-based chemotherapy regimen for EC. Participants may have received up to 1 additional line of platinum-based chemotherapy if given in the neoadjuvant or adjuvant setting and must not have received prior therapy with an ICI or other immunotherapy.

### Cohort D (MSS mCRC, IO Naïve):

Patients must have histologically or cytologically confirmed, advanced or metastatic, unresectable adenocarcinoma of the colon or rectum. All other histological types are excluded

Patients must have failed 2 lines of standard chemotherapies, including fluorouracil, oxaliplatin, and irinotecan. Failed chemotherapies are defined as the occurrence of PD or intolerable toxicities during the treatment or after the last dose.

Notes: a) Each line of treatment for advanced disease until PD includes one or more chemotherapy drugs used for ≥ 1 cycle; b) Previous adjuvant/neoadjuvant therapy is allowed. If relapse or metastasis occur during the adjuvant/neoadjuvant treatment period or within 6 months after the completion of the above treatment, that adjuvant/neoadjuvant therapy is considered as the failure of first line systemic chemotherapy for PD.

Patients with RAS wild-type tumor must have received anti-VEGF and/or endothelial growth factor receptor (EGFR) antibody treatment. Patients with RAS mutation or RAS status unknown must have received anti-VEGF antibody treatment.

Tumor tissue must have been assessed for MSS status prior to enrollment. The results should be available in the source documents and be those used to make treatment decisions for the patient. A redacted copy of the local results should accompany the archival tumor samples submitted as part of the protocol.

### Overall study conduct

In all parts of the study, there is no predefined duration of treatment for each patient. That is, patients will continue receiving study drug administration until radiologically determined PD per RECIST v 1.1, unacceptable toxicity, death, or withdrawal from study.

Treatment cycles will occur consecutively without interruption, except when necessary to manage toxicities or for administrative reasons.

The dose for fruquintinib can be reduced at any time due to the intolerable toxicity following the DLT observation window in the safety lead-in phase. Once reduced, the dose cannot be re-escalated to the previous level. There is no dose reduction for tislelizumab in this study.

The investigator has the right to discontinue a patient from the study for any condition that the investigator determines is in the best interest of the patient, any reasons of non-compliance (eg, missed doses and visits), or pregnancy.

Any patient who discontinues treatment is protocol-required to return to the study site for an EOT (end of treatment) visit and safety follow-up visit.

The EOT (end of treatment) visit is conducted  $\leq 7$  days ( $\pm 3$  days) after the last dose when the investigator determines that the patient must permanently discontinue all study drugs.

Patients who permanently discontinue all study drugs will be asked to return to the clinic for the safety follow-up visit, which is required to be conducted 30 days ( $\pm 7$  days) after the EOT visit.

Every 8 weeks (±14 days) after the EOT visit, the investigator or their designee should call the patients to collect information related to survival status and their use of other anticancer treatments, including drug name, dosage, and treatment start and end dates.

The end of the study is defined as the last visit of the last patient in the study.

The SRC will review the data during Part 2 on an ongoing basis for safety.

The study scheduled assessments are presented in Appendix 1.

# 2.3. Determination of Sample Size

Approximately 146 to 152 patients are estimated to be enrolled in this study (approximately 6 to 12 patients in the dose escalation phase and approximately 140 patients in the dose expansion phase).

### Safety Lead-In Phase

Approximately 6 to 12 patients will be enrolled into this phase of the study. The total sample size will be determined by the incidence of DLTs in the safety lead-in phase.

### Dose Expansion Phase

Approximately 30 patients will be enrolled in each of the Cohorts A and B, approximately 40 patients in Cohort C, and approximately 40 patients in Cohort D in the dose expansion phase of the study. Planned patient enrollment for each cohort can provide adequate precision for the estimate of ORR at a specific time point.

Table 1 Shows the range of ORR and the corresponding 95% CIs for a sample size of 30 or 40 patients.

Table 1 Estimated ORR and 2-Sided 95% Confidence Intervals

| Number of patients | Number of<br>Responders | Estimated ORR | 95% CI Lower<br>Limit | 95% CI<br>Upper Limit |
|---|---|---|---|---|
| 30 | 0 | 0.00 | 0.00 | 0.12 |
| 30 | 5 | 0.17 | 0.06 | 0.35 |
| 30 | 10 | 0.33 | 0.17 | 0.53 |
| 30 | 15 | 0.50 | 0.31 | 0.69 |
| 30 | 20 | 0.67 | 0.47 | 0.83 |
| 30 | 25 | 0.83 | 0.65 | 0.94 |
| 30 | 30 | 1.00 | 0.88 | 1.00 |
| 40 | 0 | 0.00 | 0.00 | 0.09 |
| 40 | 5 | 0.13 | 0.04 | 0.27 |
| 40 | 10 | 0.25 | 0.13 | 0.41 |
| 40 | 15 | 0.38 | 0.23 | 0.54 |
| 40 | 20 | 0.50 | 0.34 | 0.66 |
| 40 | 25 | 0.63 | 0.46 | 0.77 |
| 40 | 30 | 0.75 | 0.59 | 0.87 |
| 40 | 35 | 0.88 | 0.73 | 0.96 |
| 40 | 40 | 1.00 | 0.91 | 1.00 |

CI=confidence interval; ORR=objective response rate 95% Clopper-Pearson interval for binomial distribution

#### 3. ANALYSIS SETS

## 3.1. Definition of Analysis Sets

#### 3.1.1. Enrolled Set

The enrolled set includes all patients who have signed ICF (inform consent form).

### 3.1.2. Safety Analysis Set

The safety analysis set includes all enrolled patients who received at least one dose of fruquintinib or tislelizumab. The safety evaluation will be performed based on the first dose of study treatment received by a patient. This is the primary population for safety and efficacy analyses.

# 3.1.3. DLT-Evaluable Analysis Set

The DLT-evaluable analysis set included all patients enrolled in the Safety Lead-in portion of the study who received at least 1 dose of fruquintinib or tislelizumab and were considered DLT evaluable based on the SRC review, according to the pre-specified criteria from the protocol.

### 3.1.4. Response Evaluable Analysis Set

The response evaluable analysis set will include all patients who are in the safety analysis set and have a baseline tumor assessment, and either (i) have had at least one post-baseline tumor assessment, or (ii) do not have post-dose tumor assessment but have clinical progression as noted by the investigator or have died due to disease progression before their first post-baseline tumor scan. Sensitivity analysis for efficacy endpoints ORR, DCR, and CBR will be conducted using this analysis set.

### 3.1.5. Pharmacokinetics (PK) Analysis Set

The pharmacokinetic analysis set includes all patients in the safety analysis set that have at least one quantifiable plasma concentration of fruquintinib and/or tislelizumab.

### 3.1.6. Antidrug Antibody (ADA) Analysis Set

The antidrug antibody analysis set includes all patients who received at least one dose of tislelizumab and have a baseline and at least one post-baseline ADA result.

#### 3.2. Protocol Deviation

Protocol deviations including deviations that are related to COVID-19 are recorded in the Clinical Trial Management System as outlined in the latest version of the Protocol Deviation and Non-compliance Management Plan. Protocol deviations are categorized as major/minor before database lock. Certain protocol deviations are major in that they may affect the ability to assess the safety and efficacy of study drug.

#### 4. ENDPOINTS

## 4.1. General Principles for Derived and Transformed Data

### 4.1.1. Reference Start Date and End Date and Study Day

Reference start date is defined as the first date when a non-zero dose of any study drug (i.e. fruquintinib or tislelizumab, whichever occurs first) was administrated (first administration/dose date). Day 1 is the day of the first dose of study treatment in Cycle 1.

Study Day will be calculated from the reference start date, and it will be used to show start/stop day of assessments and events relative to the first administration of study treatment.

- If the date of the event is on or after the reference start date, Study Day = (date of event reference start date) + 1.
- If the date of the event is prior to the reference start date, Study Day = (date of event reference start date).

In the situation where the event date is partial or missing, the date will appear partial or missing in the listings.

Reference end date is defined as the last date when a non-zero dose of any study drug was administered

### 4.1.2. Baseline and Change from Baseline

Baseline is defined as the last non-missing assessment prior to the first administration of any study drug (whichever occurs first), including scheduled and unscheduled visits, unless otherwise specified. For quantitative measurements:

- change from baseline (CFB) will be calculated as: CFB = Assessment value at visit X –
  Baseline value;
- percentage CFB (% CFB) will be calculated as % CFB = (Assessment value at each visit X Baseline value)/Baseline value × 100.

#### 4.1.3. Treatment Period

Unless otherwise specified, the treatment period is defined as the period from first administration date to [30 days + 7 days protocol defined window] after last administration date on treatment. For safety data, only the assessments/events collected during the treatment period will be evaluated (except for related SAE and immune-mediated AE [imAEs]).

The worst post baseline is defined as the worst assessments/events during the treatment period including both scheduled and non-scheduled visits. The last assessment on treatment measurement is defined as the latest non-missing measurement taken during the treatment period.

# 4.2. Efficacy Endpoints

## 4.2.1. Primary Endpoint

The primary efficacy endpoint for Part 2 is the objective response rate (ORR) which is defined as the proportion of patients with a confirmed best overall response (BOR) complete response (CR) or Partial Response (PR) as determined by the investigator using RECIST v1.1.

BOR will be determined using time point responses (TPRs) up until the last evaluable TPR prior to or on the date of (i) disease progression as defined by RECIST Version 1.1 (Eisenhauer 2009) or death; or (ii) withdrawal of consent or lost to follow-up; or (iii) receiving subsequent anti-cancer therapy (i.e. medication, not including the radiotherapy and procedure), whichever is earlier.

The timing of an overall TPR will always be derived based on scan dates not response assessment dates. For a scheduled tumor scan assessment, it is expected that there may be a variation for the actual timing of scans among target, non-target, and new lesions. In assigning a date for the overall response assessment at a visit, the earliest date collected at that visit will be used. Within a grouped timepoint, if there are multiple assessments on different dates for the same target lesions, the last assessment will be used.

A patient's BOR will be determined based on Table 2.

There are two ways of assigning BOR for a patient when the minimum interval for confirmation of CR and PR is not satisfied or if there are no confirmatory scans for CR and PR:

- Adding two more response categories as: unconfirmed CR, unconfirmed PR;
- Assigning BOR as SD, that is, both the unconfirmed CR and unconfirmed PR will be SD.

Both ways of assigning BOR will be implemented.

The number and percentage of patients in each category of derived BOR (Confirmed CR, Confirmed PR, SD, PD, or not evaluable]) will be summarized.

A patient who is in the safety analysis set but not in the response evaluable analysis set, or in response evaluable analysis set, but does not have any post-baseline tumor assessment (patients who died or progressed clinically prior to the first scheduled tumor assessment), the response category "NA" will be assigned for BOR of the patient.

Table 2 Best Overall Response When Confirmation of CR and PR are Required

| First TPR | Second TPR [a] | Best overall<br>response*^ for ORR | Best Overall Response for ORRUNCONFIRMED |
|---|---|---|---|
| CR | CR | CR | CR |
| CR | PR | SD [b] or PD | Unconfirmed CR |
| CR | SD | SD [b] or PD | Unconfirmed CR |
| CR | PD | SD [b] or PD | Unconfirmed CR |
| CR | NE or NA | SD [c] or NE or NA | Unconfirmed CR |
| PR | CR | PR | Unconfirmed CR |
| PR | PR | PR | PR |

| PR | SD | SD [d] | Unconfirmed PR |
|----------|------------|--------------------|----------------|
| PR | PD | SD [b] or PD | Unconfirmed PR |
| PR | NE or NA | SD [c] or NE or NA | Unconfirmed PR |
| NE | NE | NE | NE |
| NE | CR | SD | Unconfirmed CR |
| NE | PR | SD | Unconfirmed PR |
| NE | SD | SD | SD |
| NE or NA | PD | PD | PD |
| SD | PD | SD [b] or PD | SD [b] or PD |
| SD | CR | SD | SD |
| SD | PR | SD | SD |
| SD | SD | SD | SD |
| SD | NE or NA | SD [c] or NE or NA | SD [c] or NE |
| PD | No further | | |
| | evaluation | PD | PD |

CR = Complete Response; NE = Not Evaluable; NA = Not Available; ORR = Objective Response Rate; PD = Progressive Disease; PR= Partial Response; SD = Stable Disease.

### 4.2.2. Secondary Endpoints

### 4.2.2.1. Progression-free Survival (PFS)

Progression-free survival (PFS) is defined as the time (months) from start of study treatment (fruquintinib or tislelizumab) until the first radiographic documentation of objective progression as assessed by the investigator using RECIST v1.1, or death from any cause.

More specifically, PFS will be determined using all the assessment data up until the last evaluable visit prior to or on the date of:

- disease progression as defined by RECIST Version 1.1 or death; or
- (ii) withdrawal of consent or lost to follow-up; or
- (iii) receipt of subsequent anti-cancer therapy (i.e. medication, not including the radiotherapy and procedure), whichever is earlier.

<sup>[</sup>a] The minimum interval for confirmation of CR and PR is 4 weeks.

<sup>[</sup>b] Best response will be SD if the first time point overall response is after 49 days (8 weeks from start of treatment and allowing a 7 day visit window) on study. Otherwise, the best response will be PD.

<sup>[</sup>c] Best response will be SD if the first time point overall response if after 49 days on study. Otherwise, the best response will be NE.

<sup>[</sup>d] Best response will be SD provided the criteria for PD have not been met from the first to second assessment.

<sup>\*</sup> A best overall response of SD can only be made after the patient is on study for a minimum of 49 days (counted from Cycle 1 Day 1). If the patient is on study for less than 49 days, any tumor assessment indicating stable disease before this time period will have a best response of NE unless PD is identified.

<sup>^</sup> Subsequent documentation of a CR may provide confirmation of a previously identified CR even with an intervening NE (e.g., CR NE CR). Subsequent documentation of a PR may provide confirmation of a previously identified PR even with an intervening NE or SD (e.g., PR NE PR or PR SD PR). However, only one (1) intervening NE or SD will be allowed between PRs for confirmation. Note: in the following scenario, PR SD NE PR, the second PR is not a confirmation of the first PR.

Patients without report of PD or death from any cause at the time of analysis are censored as described in Table 3 below.

The PFS time will always be derived based on scan dates not tumor assessment dates. RECIST assessments/scans contributing towards a particular visit may be performed on different dates. The following rules are applied:

- Date of progression is determined based on the earliest of the dates of the component that triggered the progression.
- When censoring a patient for PFS, the patient is censored at the latest of the dates contributing to a particular overall visit assessment.

Table 3 Censoring Rules for PFS

| Rule | Situation | Date of Progression or Censoring | Outcome |
|---|---|---|---|
| 1 | PD documented from radiological assessment visits | Date of documented disease progression | Event |
| 2 | Death without PD or death before first<br>documented PD or death after one<br>missing radiological assessment visit | Date of death | Event |
| 3 | No baseline or post-baseline radiological assessments available | Date of start of study treatment | Censored |
| 4 | No death or PD by the time of data cut-off for final analysis | Date of last adequate radiological assessment | Censored |
| 5 | Early discontinuation (lost to follow-<br>up or withdrawal of consent) of study<br>without death or PD | Date of last adequate radiological assessment | Censored |
| 6 | New anti-tumor medication started prior to PD or death | Date of last adequate radiological assessment prior to or on date of initiation of new medication visit. In case of no post-baseline tumor assessments, it will be the date of first study treatment administration | Censored |
| 7 | Death or PD occurred after two or<br>more consecutive missed radiological<br>assessment visits | Date of last adequate radiological assessment prior<br>to missed visits. In case of no post-baseline tumor<br>assessments, it will be the date of first study<br>treatment administration | Censored |

Note: An adequate radiologic assessment is defined as an assessment where the Investigator determined radiological response is CR, PR, SD, or PD. If PD and new anti-cancer therapy occur on the same day, will assume that the progression was documented first, e.g. outcome is progression and the date is the date of the assessment of progression

Note: Two consecutive scheduled tumor assessments is equal to 126 days (=2\* (8 weeks \*7+ 7 days)) since previous evaluable RECIST 1.1 or baseline assessment if there is no post baseline tumor assessment.

#### 4.2.2.2. Disease Control Rate

Disease control rate (DCR) is defined as the proportion of patients with a BOR of CR, PR, or SD lasting for at least 7 weeks as determined by the investigator using RECIST v1.1. A patient who is in the safety analysis set but not in response evaluable analysis set, or in response

evaluable analysis set, but does not have any post-baseline tumor assessment (patients who died or progressed clinically prior to the first scheduled tumor assessment), the response category "No" will be assigned for DCR of the patient.

#### 4.2.2.3. Clinical Benefit Rate

Study Protocol: 2020-013-00US3

Clinical benefit rate (CBR) is defined as the proportion of patients with a BOR of CR, PR, or durable SD (i.e. lasting for at least 6 months) as determined by the investigator using RECIST v1.1. A patient who is in the safety analysis set but not in response evaluable analysis set, or in response evaluable analysis set, but does not have any post-baseline tumor assessment (patients who died or progressed clinically prior to the first scheduled tumor assessment), the response category "No" will be assigned for CBR of the patient.

## 4.2.2.4. Duration of Response

Duration of response (DoR) is defined as the time from the first occurrence of PR or CR by RECIST Version 1.1, until disease progression or death, whichever comes first.

Only those patients with confirmed objective responses of CR or PR will be included in this analysis.

Censoring will follow the rules outlined for PFS in Table 3 of Section 4.2.2.1.

For those patients with confirmed objective responses of CR or PR, DoR is calculated as (date of death or PD or last assessment – date of first occurrence of CR or PR + 1)/30.4375.

#### 4.2.2.5. Overall Survival

Overall survival is defined as the time (months) from the start of study treatment (fruquintinib or tislelizumab) until the date of death due to any cause.

That is, OS will be calculated as (date of death or last known alive – date of start of study treatment + 1)/30.4375.

In rare case, if year and month of death date are known but the day is unknown, day will be imputed as 15. For example, if a patient is reported to die on Dec2017, the death date will be imputed as 15 Dec2017. In the case of the imputed death date being after the end of study date and the death date and end of study date being the same month, the death date will be assigned to be the date of end of study.

Patients with no event during the study will be censored at the date last known to be alive. OS will not be censored if a patient receives subsequent anticancer treatments after discontinuation of the study drugs.

Moreover, the last known alive date will be derived for patients not known to have died at the analysis cut-off date using the latest date (including complete date and partial date with Month and Year information) among the following data:

 All assessment dates (e.g. laboratory, vital signs assessments, ECG, ECOG, performance status assessment, tumor assessment dates etc.).

- Medication dates including study medication, concomitant medications, anticancer therapies administered after study treatment discontinuation.
- Adverse events start and end date.
- Date latest known alive collected during the survival follow-up.

After sorting properly for all those available dates, if the last known alive date is a partial date with Month and Year information, day will be imputed as 15, unless this is after the cut off date in which case the cutoff date will be used as last alive date.

# 4.3. Exposure Endpoints

Drug exposure, including number of cycles received, total duration of exposure, cumulative dose received (mg), dose intensity, and relative dose intensity of fruquintinib and tislelizumab will be calculated as per algorithms included in Table 4.

The total duration of exposure (days) for fruquintinib will be calculated from the first dose date of fruquintinib in Cycle 1 to the last dose date of fruquintinib + 8 days or death date, whichever comes earlier if treatment is discontinued, or to the cut-off date if treatment is still ongoing. The total duration of exposure (days) for tislelizumab will be calculated from the first dose date of tislelizumab in Cycle 1 to the last dose date of tislelizumab + 28 days or death date, whichever comes earlier if treatment is discontinued, or to the cut-off date if treatment is still ongoing. The total duration of exposure (days) will be calculated from the first dose date of either study drug (fruquintinib or tislelizumab) in Cycle 1 to the earlier date between the last dose date of fruquintinib + 8 days and last dose date of tislelizumab + 28 days, or death date, whichever comes earlier if treatment is discontinued, or to the cut-off date if treatment is still ongoing.

### Number of Cycles Received

Patients are considered to have started a cycle if they have received at least one dose of any study drug (fruquintinib or tislelizumab). In addition to the numeric summary for the number of cycles, the number of cycles will be categorized as 1, 2, 3, 4, 5, and  $\geq 6$ .

# Total Dose Administered (mg) in a Cycle for fruquintinib

In the study, fruquintinib (at a dose of 5 mg) is provided for oral administration, and in the event of dose adjustment, 1 mg fruquintinib capsules can be used.

Based on drug accountability data, the number of capsules taken for each dose level will be calculated as total dispensed – total returned in a cycle, then, the total dose administered (mg) in a cycle will be the summation as (number of 5mg capsules taken  $\times$  5 + number of 1mg capsules taken).

Table 4 Algorithms for Calculating Parameters Relevant to the Dose Exposure and Intensity

| Parameter | Fruquintinib § | Tislelizumab |
|---|---|---|
| Dosing Schedule | 5 mg PO QD (3 weeks on/1 week off) | 300 mg IV on Day 1 of a 4- |
| per Protocol | | weeks cycle |
| Number of Cycles | Patients will be considered to have star | |
| Treatment | at least one dose of study drugs (frug | - |
| Received | respective of | cycle. |
| Dose by cycle | Total dose administered (mg) | Total dose administered (mg) |
| Cumulative Dose | Sum of the doses administered to a pa | tient in the duration of exposure |
| (mg) | (mg) | |
| Dose intensity | Cumulative dose (mg) / (duration of exposure) (day) | |
| (mg/day) | , ,, | * / / */ |
| Relative dose | 100 * [Dose intensity (mg/day) / (5 | 100 * [Dose intensity (mg/day) |
| intensity (RDI) (%) | *21 /28 (mg)] | / (300 /28 ] |
| | 100 * [Cumulative dose (mg) / | 100 * [Cumulative dose (mg) / |
| Relative dose (%) | $(5\times21\times number of cycles for$ | (300 × number of cycles for |
| | fruquintinib (mg)] | tislelizumab (mg)] |
| Number of Days | | |
| with any recorded | Sum of days with recorded doses | NA |
| dose | | |
| Percentage | 100 * [(number of days with any | |
| Intended Dose | recorded doses)/duration of | NA |
| (PID) (%) | exposure], target PID is 75%. | |

<sup>§</sup> Two different doses (5 mg PO QD and 4 mg PO QD) of fruquintinib may be evaluated in Part 1. The 5 mg PO QD is expected to be the planned dose for patients in Part 2. The calculation of relevant parameters will be adjusted accordingly based on the example presented in this table.

 $PO = Per \ os \ (oral \ administration); QD = Quaque \ die \ (once \ daily).$ 

In addition, the RDI (%) and RD (%) will be categorized to the groups: < 50%; 50 - < 70%; 70 - < 90%; 90 - < 110%;  $\ge 110\%$ .

### Study Drug Adjustment

The following endpoints to reflect study drug adjustment in the duration of exposure will be derived. Dose reduction is not allowed for tislelizumab.

- <u>Dosing modifications</u> (including both dosing interruption and dose reduction): number of patients with any dosing modification, and categorized frequency of dosing modification (0, 1, 2, 3, 4, > 4). This will be derived only for fruquintinib.
- <u>Dosing interruption</u>: number of patients with any dosing interruption and reasons for dosing interruption, and categorized frequency of dosing interruptions (0, 1, 2, > 2).

 Date: 29 July 2024

 <u>Dose reduction</u>: number of patients with any dose reduction and reasons for dose reduction, and categorized frequency of dose reduction (0, 1, 2, > 2). This will be derived only for fruquintinib.

## 4.4. Safety Endpoints

The safety analysis set is used to evaluate the safety variables including adverse events, clinical laboratory data, vital signs, single 12-lead ECG parameters, ECHO/MUGA parameters, physical examinations, ECOG performance status, and death. The safety data during the treatment period will be evaluated, and the treatment period is defined as the duration from the date of the first study drug administration until [30 days + 7 days protocol defined window] after the last study drug (fruquintinib or tislelizumab) administration or the date of death, whichever comes first.

### 4.4.1. Dose Limiting Toxicities (DLTs) or DLT-equivalent

AEs will be assessed per the DLT criteria, for patients from part 1, during the 28-day DLT assessment window in Cycle 1, which starts with the first day of administration of study drugs. Moreover, for patients from Part 1, after the 28-day DLT evaluation window of Cycle 1, an AE will also be evaluated for DLT-equivalent according to the DLT criteria. Hence, an AE will be determined whether it is a DLT/DLT-equivalent or not.

## 4.4.2. Adverse Events (AEs)

All AEs will be coded from verbatim text to preferred term (PTs) and grouped by system organ class (SOC) using the MedDRA (Medical Dictionary for Regulatory Activities) Version 25.0 or higher. AEs will be collected from the time of signature of informed consent throughout the treatment period. AEs will be graded by investigator according to CTCAE, Version 5.0, missing severity grade is imputed as Grade 3.

An AE is considered a TEAE based on the following definition:

- During the treatment period from the date of the first study drug administration until 37 days after the last study drug (fruquintinib or tislelizumab) administration:
  - 1.1 if the onset date is on or after the start of study treatment (fruquintinib or tislelizumab); or
  - 1.2 if the AE has an onset date before the start of study treatment but worsened in severity;
- 2. After the treatment period regardless of whether or not the patient starts a new anticancer therapy, that is, at 37 days after the last dose of study drug (fruquintinib or tislelizumab) administration:
  - 2.1 treatment-related SAEs; or
  - 2.2 immune-mediated AEs (imAEs) recorded up to 90 days after the last dose of tislelizumab.

Other AE variables include drug-related AEs, AEs leading to study drug modifications (i.e. dose interruption, dose reduction, or study drug withdrawal), AEs leading to death, and SAEs.

An AE is considered treatment-related to fruquintinib or tislelizumab in the summaries if it is assessed as related to fruquintinib or tislelizumab by the investigator or if the assessment of relationship to study treatment is missing.

For AEs which are not ongoing, duration of AE (days) is defined as AE end date – AE start date +1; for ongoing AEs, the end date will be listed as 'Ongoing' and the duration of AE (days) will be approximated as ' $\geq$  date of last visit – AE start date +1'.

## AEs of special interest (AESI) for fruquintinib

According to the IB Version 13.0 (dated 08 November 2021), AESI for fruquintinib are defined to include 10 categories:

- hepatic function abnormal
- haemorrhages
- hypertension
- infections
- thyroid dysfunction
- proteinuria
- dermatological toxicity
- gastrointestinal perforation
- embolic and thrombotic events
- left ventricular ejection fraction decreased

The MedDRA terms used to define AESIs categories are listed in Table 5, for AESI categories (i.e. "haemorrhages", "hepatic function abnormal", "hypertension", "proteinuria", "thyroid dysfunction", "embolic and thrombotic events" "gastrointestinal perforation" and "left ventricular ejection fraction decreased"), the PTs to be included in these AESI categories are included in Appendix 3. These terms were selected by subjecting standardized MedDRA queries (SMQ) lists (narrow and/or broad scope depending on the category) for each category and had been used in the fruquintinib clinical development program for pharmacovigilance. The MedDRA terminology is subject to changes and modifications as medical knowledge develops. Thus, the terms within Table 5 and Appendix 3 could be updated/changed in the future.

Table 5 MedDRA Terms Used for Adverse Events of Special Interest

| AESIs Category | Search terms/strategy |
|---|---|
| Dermatological toxicity | MedDRA SOC "skin and subcutaneous tissue disorders" |
| Hypertension | MedDRA SMQ "hypertension" (narrow) |
| Thyroid dysfunction | MedDRA SMQ "thyroid dysfunction" (broad) |
| Proteinuria | MedDRA SMQ "proteinuria" (narrow) |
| Hepatic function abnormal | MedDRA SMQ "drug related hepatic disorders- |
| | comprehensive search" (narrow) |
| Haemorrhages | MedDRA SMQ "haemorrhages" (narrow) |
| Infections | MedDRA SOC "infections and infestations" |
| Embolic and thrombotic events | MedDRA SMQ "embolic and thrombotic events" (narrow) |

| AESIs Category | Search terms/strategy |
|---|---|
| Gastrointestinal perforation | MedDRA SMQ "gastrointestinal perforation" (narrow) |
| Left ventricular ejection fraction | MedDRA SMQ "cardiac failure" (narrow) |
| decreased | |

Time to first AESI is defined as time interval from date of first administration of study drug (fruquintinib/tislelizumab) to the earliest onset date among TEAEs within the same AESI categories. That is, if a patient has multiple AEs occurrences under the same AESI category, the earliest AE onset date will be used as the first onset date to the AESI category.

## Immune-mediated AEs (imAE)

Immune mediated AEs will be identified based on the AE standardized MedDRA queries (SMQs). imAEs categories are immune-mediated AEs, serious skin adverse reactions and diabetes. The PTs to be included in these imAEs categories are included in Appendix 4.

#### COVID-19 Related AE

COVID-19 related AE will be identified based on the preferred term list (MedDRA version 25.0) included in <u>Appendix 5</u>.

### 4.4.3. Laboratory

Blood and urine samples for the determination of clinical chemistry, hematology, and urinalysis laboratory variables described in Table 6 will be measured.

Table 6 Laboratory Assessment

| Lab Category | Lab tests |
|---|---|
| Hematology | Red blood cell count, hemoglobin, hematocrit, reticulocyte count, white |
| | blood cell count and classifications (neutrophils, lymphocytes, eosinophils, |
| | monocytes, and basophils), and platelet count |
| Chemistry | Albumin, blood urea nitrogen or urea, creatinine, CrCl rate, ALT, AST, |
| | alkaline phosphatase (ALP), bicarbonate, non-fasting total cholesterol, |
| | triglycerides, uric acid, lactate dehydrogenase, bilirubin/total bilirubin, |
| | Urea, sodium, potassium, magnesium, chloride, glucose, corrected calcium |
| | (for patients with hypoproteinemia), total protein, phosphorus, blood |
| | glucose, creatine phosphokinase, creatine kinase-MB (CK-MB), amylase |
| | and lipase |
| | If CK-MB fractionation is not available, troponin I and/or troponin T |
| | should be tested instead |
| Fasting Lipid | Total cholesterol, High-density lipoprotein, Low-density lipoprotein, |
| Panel | Triglycerides |
| Coagulation | Prothrombin time, INR, and aPTT |

 Lab Category
 Lab tests

 Thyroid
 Serum free tri-iodothyronine (FT3), serum free thyroxine (FT4), and thyroid stimulating hormone (TSH).

 Urinalysis
 Urine pH, protein, glucose, white blood cell, red blood cell

Change from baseline in laboratory test results to each assessment will be calculated.

The non-protocol specified tests (if any reported) and urinalysis results will not be summarized; they will only be included in listings.

Data recorded by the laboratory will be converted to the International System of Units (SI) and all presentations will use SI units.

Quantitative laboratory measurements reported as "< X", i.e. below the lower limit of quantification (LLQ), or "> X", i.e. above the upper limit of quantification (ULQ), will be converted to X for the purpose of quantitative summaries, but will be presented as recorded, i.e. as "< X" or "> X" in the listings.

Clinical laboratory results will be graded according to CTCAE criteria, CTCAE v5.0 criteria (see Appendix 2). Any graded abnormality that occurs following the initiation of study drug and represents at least a 1-grade increase from the baseline assessment is defined as treatment emergent. Any assessment for which CTCAE toxicity grades are not available will not be included in any analyses for which toxicity grades are required.

For the urinalysis parameters, if the test result is "-" or "negative", the investigation interpretation for the lab test will be considered to be "normal". The information of converting urinalysis parameters (i.e. WBC, RBC, and protein) results is provided in <u>Appendix 6</u>.

### Analysis of Abnormal Hepatic Laboratory Values

The following categories of abnormal hepatic laboratory values will be evaluated for any occurrence among all post baseline assessments.

- Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3x upper limit of normal (ULN) and ≤ 5x ULN
- AST > 3,5,8,10, and 20x ULN, AST>5x ULN for more than 5 weeks
- ALT > 3,5,8,10, and 20x ULN, ALT > 5x ULN for more than 5 weeks
- AST and/or ALT > 3,5,8,10, and 20x ULN, >5x ULN for more than 5 weeks
- Total bilirubin elevations > 1.5x, 2x ULN
- ALP > 1.5x, 2x ULN
- POTENTIAL DRUG-INDUCED LIVER INJURY (DILI): AST and/or ALT > 3x ULN and total bilirubin > 1.5x, > 2x ULN)
- AST and/or ALT >3x ULN and (total bilirubin > 2x ULN or INR > 1.5)

Hy's Law criteria: AST and/or ALT > 3x ULN and total bilirubin ≥ 2x ULN and ALP < 2x ULN</li>

Additionally, the last assessment on treatment, minimum, maximum values for each patient over the entire treatment period for each hematology and chemistry laboratory parameter will also be derived. The change from baseline will be calculated using these minimum and maximum values.

### 4.4.4. ECG

Electrocardiogram (ECG) parameters include heart rate, PR interval, RR interval, QT, QTcF and QRS intervals. Change from baseline to each post-baseline visit will be calculated and summarized by visit.

Potentially clinically significant ECG findings will be identified using the criteria which are included in Table 7.

Additionally, the last assessment on treatment, minimum and maximum values for each patient over the entire treatment period for each ECG parameter will also be derived. The change from baseline will be calculated using these minimum and maximum values.

Table 7 Potentially Clinically Significant Criteria for ECG

| ECG Parameter (unit) | Criterion value |
|----------------------|---------------------------------------|
| Heart Rate (bpm) | >120 |
| ``` | <50 |
| PR Interval (ms) | ≥ 210 |
| RR Interval (ms) | > 1200 |
| | < 500 |
| QRS Interval (ms) | ≥ 120 |
| | ≤ 50 |
| QT Interval (ms) | ≥ 500 |
| | ≤300 |
| QTcF (msec) | > 450 |
| | > 480 |
| | > 500 |
| | ≤ 300 |
| | Increase from baseline > 30 |
| | Increase from baseline > 60 |
| | > 450 and increase from baseline > 30 |
| | > 450 and increase from baseline > 60 |
| | > 480 and increase from baseline > 30 |

| > 480 and increase from baseline > 60 |
|---------------------------------------|
| > 500 and increase from baseline > 30 |
| > 500 and increase from baseline > 60 |

# 4.4.5. Vital Signs

Vital signs include systolic blood pressure (SBP), diastolic blood pressure (DBP), respiratory rate, heart rate, body temperature, weight, height, Body Mass Index (BMI) will be computed as weight (kg)/[height (m)]<sup>2</sup>.

For vital signs, change from baseline to each post-baseline visit and timepoint will be calculated.

Potentially clinically significant findings of vital signs will also be defined based on criteria in Table 8.

Additionally, the last assessment on treatment, minimum and maximum values for each patient over the entire treatment period for each vital sign parameter will also be derived. The change from baseline will be calculated using these minimum and maximum values.

Table 8 Potentially Clinically Significant Criteria for Vital Signs

| Vital Sign Parameter | Criterion value |
|--------------------------|--------------------------------------|
| | Increase from baseline of |
| | > 0 - ≤ 20 |
| SBP (mmHg), DBP | > 20 - ≤ 40 |
| (mmHg), Heart rate (bpm) | > 40 |
| Respiratory rate | Decrease from baseline of |
| (breaths/min) | > 0 - ≤ 20 |
| | > 20 - ≤ 40 |
| | > 40 |
| | Percentage decrease from baseline of |
| | < 5% |
| | ≥ 5 − < 10% |
| | ≥ 10 - < 20% |
| Weight (Ira) | ≥ 20% |
| Weight (kg) | Percentage increase from baseline of |
| | < 5% |
| | $\geq 5 - < 10\%$ |
| | ≥ 10 - < 20% |
| | ≥ 20% |

#### 4.4.6. Performance Status

Eastern Cooperative Oncology Group (ECOG) performance status is collected at screening, during the treatment period (i.e. Day 1 of each Cycle), at EOT and follow-up.

### 4.4.7. Echocardiogram

ECHOs will be done at Screening and every 12 weeks from C1D1 thereafter through the end of treatment visit. Assessment parameters include left ventricular ejection fraction (LVEF) and overall interpretation of cardiac function. Multiple-gated acquisition scans (MUGAs) are permitted if ECHOs cannot be performed.

### 4.4.8. Physical Examination

A comprehensive physical examination (PE) at Screening, it includes general appearance, eyes, ears, nose and throat, head and neck, respiratory, cardiovascular, abdomen (gastrointestinal), skin, genitourinary system, lymph nodes, musculoskeletal, neurological assessments.

Limited physical examination at scheduled visits is a subset the comprehensive physical examination as deemed appropriate by the investigator.

Abnormal clinically significant findings in PE were to be reported as AEs (post-baseline) or MHs (screening).

These data will only be available in listings.

## 4.5. Other Endpoints

# 4.5.1. Pharmacokinetic Endpoint

Blood samples will be collected for analysis of fruquintinib and metabolite M11 plasma concentrations and tislelizumab serum concentrations according to the PK schedule of events in Table 2 of the protocol.

### 4.5.2. Immunogenicity

Serum samples will be collected for antidrug antibody (ADA) analysis to tislelizumab according to the PK schedule of events in Table 2 of the protocol.

## 4.5.3. Exploratory Endpoints

Distribution of PD-L1 expression or MSS/MSI status will be examined in all patients. Other potential predictive markers including, but not limited to, TILs, TMB, cytokine expression, and gene signature profiling may be detected and analyzed.

#### 5. ANALYSIS METHODS

# 5.1. General Principles

## 5.1.1. General Methodology

In general, all efficacy and safety will be summarized using descriptive statistics and graphs as appropriate. Continuous variables will be summarized by descriptive statistics (sample size (n), mean, standard deviation, minimum, 25% percentile (Q1), median, 75% percentile (Q3), and maximum). Categorical variables will be summarized in frequency tables (frequencies and percentages).

Time to event variable will be analyzed using Kaplan-Meier method and summarized with median, 25% and 75% percentiles with their corresponding 95% confidence intervals (CI) which are calculated from a log-log transformation based on the method by Brookmeyer 1982

. Individual data will be presented in patient listings which will be provided for all patients.

Analyses will be implemented using SAS® 9.4 or higher (SAS Institute, Cary, North Carolina, USA). The International Conference on Harmonization (ICH) numbering convention, i.e. ICH-E3, will be used for all tables and listings.

All summary tables, listings, and figures (TLFs) will be presented by cohorts as defined in Table 9. Unless otherwise specified, for Cohort A and Cohort B, the TLFs will be presented overall, by cohort, and by category of ER/PR positivity per ASCO-CAP guidelines (Allison 2020). TNBC will be defined as ER/PR positivity of <1%, and ER/PR low positive disease will be defined by ER/PR positivity of 1% to 10%. If a patient from Part 1 has the same type of cancer evaluated in Part 2, the patient from Part 1 will also be included in relevant group for analysis in Part 2.

Table 9 Treatment/Cohort Display in TLFs

| Part of the study | Group | Group Description in Data<br>Display | Subgroup |
|---|---|---|---|
| Part 1 | 1 | Fruquintinib 5 mg +<br>Tislelizumab | NA |
| | 2† | Fruquintinib 4 mg +<br>Tislelizumab | NA |
| Part 2 [a] | 1 | Cohort A BC (IO-Treated) | TNBC |
| | | | ER/PGR low positive |
| | | | Total |
| | 2 | Cohort B BC (IO-Naïve) | TNBC |
| | | | ER/PGR low positive |
| | | | Total |
| | 3 | Cohort C endometrial | NA |
| | | cancer | |

 Date: 29 July 2024

| Part of the study | Group | Group Description in Data<br>Display | Subgroup |
|-------------------|-------|--------------------------------------|----------|
| | 4 | Cohort D MSS mCRC (IO<br>Naïve) | NA |

<sup>†</sup> this cohort may not be explored in the conduct depending on observed toxicity from the dose cohort 5 mg PO QD ER/PGR: receptor/progesterone receptor

For continuous data, unless otherwise specified, the mean, median, Q1, and Q3 will be presented with one more significant digit than the original values, and standard deviation will be reported with 2 more significant digits than the original values. The minimum and maximum should report the same significant digits as the original values. The derived variables will be presented with one decimal place. Percentages will be reported with one decimal point; if the count is 0, no percentage will be presented. Value of percentage less than 1% will be presented as "<1%." Value of percentage less than 100% but ≥ 99.5% will be presented as ">99%." Any rounding will be done after all calculations are made.

### 5.1.2. Handling Missing Data

In general, the observed case (OC) data for a visit will consist of the actual observations recorded for the visit. If missing, the OC data will remain missing — no missing imputation will be performed. Safety analyses will be conducted on the OC data only.

However, imputation of missing AE and concomitant medication onset and stop dates will be used to determine the status of each AE and the prior/concomitant status of each medication. The specific imputation rules are provided below, refer to Section 5.1.2.1 for the method of imputation of missing AE onset and stop date and Section 5.1.2.2 for the method of imputation of missing concomitant onset and stop dates. However, the imputed dates should not be shown in listings.

For demographic and baseline characteristics, each variable will be analyzed and/or summarized using the available data. Unless otherwise specified, patients with missing data will be excluded only from analyses for which data are not available.

#### 5.1.2.1. Adverse Events Start/End Date

AEs with onset/end dates that are partially/completely missing will be imputed as follows.

#### (i) AE start date:

- If the AE onset date is completely missing, the AE start date will be imputed as the reference start date (i.e., date of first treatment).
- If the AE onset date is partial missing, then

<sup>[</sup>a] Patients with TNBC or EC enrolled in Part 1 must meet all inclusion and no exclusion criteria for the respective cohorts noted in Part 2 and will be included in relevant cohort for analysis.

- If both the year and the month are available and the year and the month are the corresponding year and month of the reference start date, then the AE start date will be imputed as the reference start date;
- If both the year and the month are available and the year and the month are not equal to the corresponding year and month of the reference start date, then the AE start date will be imputed as the 1<sup>st</sup> day of the month;
- If only the year is available and the available year is the corresponding year of the reference start date, then the AE start date will be imputed as the reference start date;
- If only the year is available, and the available year is not equal to the corresponding year
  of the reference start date, then the AE start date will be imputed as the January 1<sup>st</sup> of the
  year
- (ii) AE end date will be imputed as below for the partial date only, the imputation rules only apply when the AE is not ongoing:
- If both the year and the month are available, AE end date will be imputed as the last day of the month;
- If only the year is available, AE end date will be imputed as the December 31st of the year.

If the imputed AE end date is after the death date for patients known to be dead at end of study or cut off date, the date of the death will be used for AE end date. If the imputed AE end date is after the last known alive date for patients alive at the end of study or cut off date, the date of last known alive date will be used for AE end date.

For AE continuing at the cut-off date, the end date will not be imputed and instead will be reported as "ongoing".

## 5.1.2.2. Concomitant Medication/Procedure/Surgery Start/End Date

Concomitant Medication/Procedure/Surgery with onset/end dates that are partially/completely missing will be imputed as follows.

- start date:
- 1st day of the month will be used to impute the start date if only the day is missing
- January 1<sup>st</sup> will be used to impute the start date if both the day and month are missing
- If the date is completely missing, then the day before the reference start date will be imputed
  as the start date.
- (ii) end date:
- Last day of the month will be used to impute the end date if only the day is missing
- December 31<sup>st</sup> of the year will be used to impute the end date if both the day and month are missing
- If the date is completely missing, assign 'continuing' status to the end date

If the imputed end date is after the death date or last known alive date, the date of the death or last known alive date will be imputed as the concomitant medication/procedure/surgery end date.

#### 5.1.2.3. Subsequent Anti-Cancer Therapy Date

When a partial new anti-tumor therapy start date is reported, every effort will be made to identify the precedence relationship of starting date of new anti-tumor therapy relative to the reference end date. Below rules will be used:

- If the date is completely missing, new anti-tumor therapy date will be imputed as reference end date + 1;
- If only the day is missing, 15th day will be imputed as the new anti-tumor therapy date;
- If both the day and the month are missing, then July 1<sup>st</sup> will be imputed as the new anti-tumor therapy;

If the imputed date is earlier than reference end date, then it will be replaced with reference end date + 1, if the imputed date is later than the date of death or last known alive date, it will be replaced with the date of death or last known alive date.

#### 5.1.2.4. Primary Diagnosis Date and Metastatic Disease Diagnosis Date

When a partial date of primary diagnosis or a partial date of first metastatic disease diagnosis is reported, the below imputation rules will be used:

- If the date is completely missing, no imputation will be conducted;
- If only the day is missing, 15th day will be assigned;
- If both the day and the month are missing, then July 1st will be assigned.

Check that the imputed date is not superior or equal to the informed consent date.

#### 5.1.3. Visit Windowing

It is expected that there will be a variation between patients in the actual number of study days from the start of administration of study drug within each cycle defined as Day 1, to the dates that the scheduled visits occur. To handle this, for tables and figures where data are grouped by visit, assessments will be categorized using visit windows based on study days (relative to the Day 1 of each cycle). The visit-window mapping is described in Table 10. Visit-based summaries will be based on the windowed visits. All data, whether or not within the visit windows, will be presented in patient's listings. Describe the visit windowing practice for the analysis of safety and efficacy variable, it is recommended to keep in mind the principle that there are no gaps between two adjacent visit windows.

For windowed visits during the treatment cycles, if more than one visit occurs during a visit window, the visit closest to the scheduled day will be assigned to the windowed visit. If two visits are equidistant from the scheduled day, the later visit will be assigned to the windowed visit. If there are multiple assessments on the same day, the worst case will be used.

For a patient who prematurely discontinues the study, the premature visit will be slotted accordingly. The window for end of treatment visit will be "last dose date of last cycle + 4 days to last dose date of last cycle + 10 days" and the window for safety follow-up visit will be "Last dose date of last cycle + 11 to last dose date of last cycle + [30 days + 7 days protocol-defined window]".

Table 10 Visit Windowing

| | | C | rcle 1 | | Cyc | le 2 | Cycle 3 and onwards | Last Cycle | End of<br>treatment | Safety follow-up |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | C1D1 | C1D8 | C1D15 | C1D21<br>[b] | C2D1 | С2D15 [b] | СЗD1 [b] | CXD1 | | |
| Scheduled<br>Day [a] | 1 | 8 | 15 | 21 | 1 | 15 | 1 | 1 | | |
| ECOG | Day 1 | | | | Day -3 to<br>EOC-3 | | Day -3 to EOC-3 | Day -3 to EOC-4 | | Last dose date of last<br>cycle + 11 to last dose<br>date of last cycle + [30<br>days + 7 days protocol<br>defined window] |
| Vital Sign | Day 1 | 2 to<br>11 | 12 to<br>18 | 19 to<br>EOC-3 | Day -3 to 8 | 9 to EOC-3 | Day -3 to EOC-3 | Day -3 to EOC-4 | Last dose<br>date of last<br>cycle +4 | Last dose date of last<br>cycle + 11 to last dose<br>date of last cycle + [30<br>days + 7 days protocol<br>defined window] |
| Hematology | | 2 to<br>11 | 12 to<br>18 | 19 to<br>EOC-3 | Day -3 to 8 | 9 to EOC-3 | Day -3 to EOC-3 | Day -3 to EOC-4 | days to last<br>dose date of | - |
| Clinical<br>Chemistry | | 2 to<br>11 | 12 to<br>18 | 19 to<br>EOC-3 | Day -3 to 8 | 9 to EOC-3 | Day -3 to EOC-3 | Day -3 to EOC-4 | last cycle +<br>10 | |
| Blood amylase<br>and lipase | | 2 to<br>11 | 12 to<br>EOC-3 | | Day -3 to 8 | 9 to EOC-3 | Day -3 to EOC-3 | Day -3 to EOC-4 | | |
| Fasting lipid<br>panel | | | | | Day -3 to 3 | | Day -3 to EOC-3 | Day -3 to EOC-4 | | |
| Coagulation | | 2 to<br>11 | 12 to<br>18 | 19 to<br>EOC-3 | Day -3 to 8 | 9 to EOC-3 | Day -3 to EOC-3 | Day -3 to EOC -<br>4 | | |
| Thyroid<br>function | | | 2 to<br>EOC-3 | | Day -3 to 8 | 9 to EOC-3 | Day -3 to EOC-3 | Day -3 to EOC-4 | | |
| Urinalysis | | | | 2 to<br>EOC-3 | Day -3 to 3 | | Day -3 to EOC-3 | Day -3 to EOC-4 | | |

Study Protocol: 2020-013-00US3

| | Cycle 1 | | | Cycle 2 | | Cycle 3 and onwards | Last Cycle | End of<br>treatment | Safety follow-up | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit | C1D1 | C1D8 | C1D15 | C1D21<br>[b] | C2D1 | C2D15 [b] | C3D1 [b] | CXD1 | | |
| ECHO/MUGA | | | | | | | Day -3 to EOC-3 | Day -3 to EOC-4 | | |
| ECG | | | 2 to<br>EOC-3 | | Day -3 to 3 | | Day -3 to EOC-3 | Day -3 to EOC-4 | | Last dose date of last<br>cycle + 4 to last dose<br>date of last cycle + [30<br>days + 7 days protocol<br>defined window] |

<sup>[</sup>a] The scheduled day is relative to Day 1 of each cycle.

Note: The end date of a cycle (EOC) is defined as one day earlier than the date of Day 1 study drug administration of its next cycle. For the last cycle (where no subsequent cycle is given), the end of cycle will be defined as Day 7 relative to the last dose of the cycle.

EOC = end of cycle.

<sup>[</sup>b] If the cycle becomes the last cycle, the upper bound of the window will use EOC-4.

<sup>[</sup>c] Every 12 weeks from C1D1 (±1 week) until progression of disease.

## 5.1.4. Adjustment of Covariates

Study Protocol: 2020-013-00US3

Not applicable

#### 5.2. Analysis Methods

#### 5.2.1. Patient Disposition

Summary of study disposition will be provided by cohort as defined in Table 9 for the following:

- Number of patients who signed the informed consent
- Number of screen failures
- Reason for screen failure
- Number of patients who did not receive study treatment
- Number of patients who received study treatment
- Patients still on study treatment, if applicable
- Reason for study treatment discontinuation
- Number of patients going into survival follow-up
- Number and percentage of patients who discontinue the study
- Reason for discontinuation of the study

A separate table will be presented to show the patients included in each analysis set and summary reasons for exclusion from an analysis set.

Patient disposition and analysis sets will be also listed.

#### 5.2.2. Protocol Deviation

Protocol deviations (including COVID-19 related protocol deviations) will be summarized descriptively for patients with at least one major protocol deviation by cohort. A patient can have multiple major and/or minor deviations and will be counted once per major and/or minor deviation. The protocol deviation summary is based on the safety analysis set.

In addition, all protocol deviations including deviations that are related to COVID-19 will be provided in a by-patient listing.

#### 5.2.3. Demographic and Other Baseline Characteristics

The following demographic and other baseline characteristics will be summarized by cohort as defined in Table 9 on the safety analysis set:

- Age (years) at screening, age groups (18-65, ≥ 65 years),
- Gender, childbearing potential (female only)
- Race
- Ethnicity
- Baseline height (cm)

- Baseline weight (kg)
- Baseline BMI (kg/m²) calculated as baseline weight (kg)/ [baseline height (m)]², BMI category (<18.5, ≥18.5 and <24, ≥24 kg/m²)</li>
- Baseline ECOG status.

#### 5.2.4. Disease Characteristics

Oncology history will be summarized descriptively by cohort as defined in Table 9 for the safety analysis set for the following:

- Type of cancer at first diagnosis
- Cancer Stage at First Diagnosis (Stage 1, Stage 2, Stage 3, Stage 4)
- Primary Tumor Location at First Diagnosis
- EC Histological Classification
- TNBC Histological Classification (Invasive Ductal Carcinoma, Other)
- Non-TNBC/Non-EC Histological Classification
- Time since first diagnosis cancer (months): it is calculated as (date of first study treatment administration – date of first diagnosis of disease + 1)/30.4375.
- Time since diagnosis of metastatic disease (months): it is calculated as (date of first study treatment administration – date of diagnosis of metastasis disease + 1)/30.4375.
- Prior oncology treatments (prior anti-cancer medication, prior anti-cancer radiotherapy, prior anti-cancer procedures)

#### 5.2.5. Medical History

The conditions/diseases from medical history are those conditions/diseases that stopped prior to the study entry. Medical history will be coded to SOC and PT using MedDRA version 25.0 or higher.

The number and percentage of patients with any past medical/surgical history within each SOC and PT will be provided by cohort on the safety analysis set.

A patient will only be counted once within a particular SOC (PT) even if he/she has multiple conditions/diseases in the same SOC (PT).

Each summary will be ordered by descending order of incidence of SOC according to total column and PT within each SOC. If the frequencies tie, an alphabetic order will be applied.

#### 5.2.6. Prior and Subsequent Anti-Cancer Therapy

Prior and subsequent anti-cancer therapy, including medication, radiotherapy, and procedure or surgery, will be summarized descriptively by cohort and overall for the safety analysis set.

#### 5.2.6.1. Prior and Subsequent Anti-Cancer Medication

Prior anti-cancer medications are defined as those taken by the patient prior to the administration of study drug. Subsequent anti-cancer medications are defined as those taken by the patient after the discontinuation of the study drug.

Prior and subsequent anti-cancer medications will be coded to Anatomical Therapeutic Classification (ATC) therapeutic group (i.e., ATC Level 2) and PT using the World Health Organization Drug Dictionary (WHO-DD) version Mar 2022 or later.

The prior anti-cancer medications will be summarized by presenting the number and percentage of patients by PT and ATC. Patients taking the same medication multiple times will only be counted once for that PT or ATC. Each summary will be ordered by descending order of incidence of ATC according to total column and PT within each ATC. If the frequencies tie, an alphabetic order will be applied.

Similarly, the subsequent anti-cancer medications will be summarized.

All prior and subsequent anti-cancer medications will be presented in patient listing.

#### 5.2.6.2. Prior and Subsequent Anti-Cancer Radiotherapy

Prior anti-cancer radiotherapy is defined as those taken by the patient prior to the administration of study drug.

Subsequent anti-cancer radiotherapy is defined as those taken by the patient after the discontinuation of the study drug.

The number and percentage of patients with at least one prior anti-cancer radiotherapy will be summarized.

All prior and subsequent anti-cancer radiotherapy will be presented in patient listing.

#### 5.2.6.3. Prior and Subsequent Anti-Cancer Procedure or Surgery

Prior anti-cancer procedure or surgery are defined as those taken by the patient prior to the administration of study drug.

Subsequent anti-cancer procedures or surgery are defined as those taken by the patient after the discontinuation of the study drug.

Prior and subsequent anti-cancer procedures or surgery will be coded to SOC and PT using MedDRA version 25.0 or higher.

The prior anti-cancer procedure or surgery will be summarized by presenting the number and percentage of patients by PT and SOC. Patients taking the same medication multiple times will only be counted once for that PT or SOC.

Each summary will be ordered by descending order of incidence of SOC to total column and PT within each SOC. If the frequencies tie, an alphabetic order will be applied.

Similarly, the subsequent anti-cancer procedure or surgery will be summarized.

All prior and subsequent anti-cancer procedures or surgery will be presented in a patient listing.

#### 5.2.7. Prior and Concomitant Medications

Prior and concomitant medications (CMs) will be coded to Anatomical Therapeutic Classification (ATC) therapeutic group (i.e. ATC Level 2) and PT using the WHO-DD version Mar 2022 or higher.

Medications taken and stopped prior to the first dose of study treatment are denoted "Prior". Medications taken prior to the first dose of study treatment and continuing beyond the first dose of study treatment or those medications started on or after the first dose of study treatment but no later than 37 days after the last dose are denoted "Concomitant".

Medication with start date/time being partially or completely missing will be assumed to be concomitant if it cannot be definitely shown that the medication was not received during the treatment period.

The prior medications will be summarized by presenting the number and percentage of patients by PT and ATC. Patients taking the same medication multiple times will only be counted once for that PT or ATC. Each summary will be ordered by descending order of incidence of ATC according to total column and PT within each ATC. If the frequencies tie, an alphabetic order will be applied.

Similarly, the concomitant medications will be summarized.

All prior and concomitant medications will be presented in patient listing.

#### 5.2.8. Concomitant Procedure

Medical or surgical procedures that started after the first dose date but no later than 37 days after the last dose date are denoted "Concomitant".

Concomitant medical or surgical procedures will be classified using the MedDRA version 25.0 or higher.

The concomitant medical or surgical procedures will be summarized by presenting the number and percentage of patients by PT and SOC. Patients having the same medical or surgical procedure multiple times will only be counted once for that PT or SOC. Each summary will be ordered by descending order of incidence of SOC according to total column and PT within each SOC. If the frequencies tie, an alphabetic order will be applied.

All concomitant medical or surgical procedures will be presented in the patient listing.

#### 5.2.9. Efficacy Analyses

The safety analysis set will be used for all efficacy analysis unless otherwise specified. No formal hypothesis testing is planned for this study. Two-sided 95% confidence intervals (CIs) will be calculated in the applicable summary, unless otherwise specified.

#### 5.2.9.1. Primary Efficacy Analyses

The number and percentage of patients in each category of derived BOR (CR, PR, Unconfirmed CR, Unconfirmed PR, SD, PD, NE, or NA) will be summarized for the safety analysis set. ORR and ORRUNCONFIRMED will be summarized by cohort as defined in Table 9.

The 95% CIs of ORR and ORR<sub>UNCONFIRMED</sub> will be calculated using the Clopper-Pearson method for each cohort.

Tumor evaluation data will be presented in listings.

#### 5.2.9.2. Secondary Efficacy Analyses

For the time to event endpoints, such as PFS, OS, and DoR, the median, 25% and 75% percentile of time-to-event will be estimated using Kaplan-Meier method with their corresponding 95% CI. For PFS and OS, additionally, estimates will be provided for the survival probability along with their 95% CIs which are calculated using linear transformation (Brookmeyer 1982)

at selected landmarks, for example, at 3, 6, 9, 12, and 18 months. The Kaplan-Meier plots will be produced for PFS and OS. The duration of follow-up will be calculated descriptively using the Kaplan-Meier method.

In order to assess duration of follow-up for PFS and OS, Kaplan Meier estimates will be calculated in the same way as in their analysis, while using different censoring rule which reverses censoring indicator instead, i.e., patients who have event will be censored at the date of event. Patients who are censored will be assigned as "event".

The DCR and CBR will be analyzed in a similar way as ORR described in Section 5.2.9.1.

#### 5.2.9.3. Sensitivity Analysis for Efficacy Endpoint

A sensitivity analysis for ORR, DCR, CBR and DoR will be conducted using the response evaluable analysis set. The analysis techniques follow those described in Section 5.2.9.1.

#### 5.2.10. Exposure of Study Treatment

Exposure of study treatment described in Section 4.3 (duration of exposure, number of cycles of treatment received, cumulative dose, dose intensity and relative dose intensity for each study drug,) will be summarized by cohort as defined in Table 9.

Number of cycles received will be categorized as (1, 2, 3, 4, 5, 6, >6, and the number and percentage of patients for each category will be summarized.

The following summary for dose modification will be summarized separately for each drug (fruquintinib and tislelizumab) by cohort. Dose reduction/increase is not allowed with tislelizumab.

 Number of patients with any dose modification with fruquintinib (including both drug interruption and dose reduction, and frequency of dose modification: 0, 1, 2, 3, 4, 5, 6, >6

- Number of patients with any drug interrupted with fruquintinib or tislelizumab (number of patients experienced drug interruption and reasons for drug interruption, and frequency of drug interruptions: 0, 1, ≥ 2)
- Number of patients with any dose reduced with fruquintinib (Number of patients with any dose reduction and reasons for dose reduction; and frequency of dose reduction: 0, 1, ≥ 2).

#### 5.2.11. Safety Analyses

Safety data during the treatment period will be summarized. The treatment period is defined as the duration from the date of the first study drug administration (fruquintinib and tislelizumab) until 37 days after the last study drug administration.

#### 5.2.11.1. Dose-Limiting Toxicity (DLT)

All DLT analysis will be only performed for Part 1 based on the DLT evaluable analysis set.

In addition to summarizing the number of patients and percentage of DLTs, DLTs will be summarized by SOC, PT, and highest CTCAE grade.

DLTs will be listed.

#### 5.2.11.2. Adverse Events

An overall summary of the number and percentage of patients along with the number of adverse events for cohort will be provided for the following categories of AEs:

| Croup | Summary scope |
|---|---|
| Group | Summary scope |
| All TEAEs | <ul> <li>CTCAE Grade ≥3 AEs</li> </ul> |
| | - Fruquintinib-related AEs |
| | - Tislelizumab-related AEs |
| | <ul> <li>AEs Leading to Dose Reduction of Fruquintinib</li> </ul> |
| | - AEs Leading to Dose Interruption of Fruquintinib |
| | AEs Leading to Dose Interruption of Tislelizumab |
| | - AEs Leading to Treatment Discontinuation of Fruquintinib |
| | <ul> <li>AEs Leading to Treatment Discontinuation of Tislelizumab</li> </ul> |
| | - Treatment-related AEs Leading to Dose Reduction of Fruquintinib |
| | - Treatment-related AEs Leading to Dose Interruption of Fruquintinib |
| | Treatment-related AEs Leading to Dose Interruption of Tislelizumab |
| | Treatment-related AEs Leading to Treatment Discontinuation of |
| | Fruquintinib |
| | - Treatment-related AEs Leading to Treatment Discontinuation of |
| | Tislelizumab |
| | - AEs Leading to Death |
| Serious TEAEs | <ul> <li>CTCAE Grade ≥3 SAEs</li> </ul> |
| | - Fruquintinib-related SAEs |
| | - Tislelizumab -related SAEs |

| Group | Summary scope |
|---|---|
| | SAEs Leading to Dose Reduction of Fruquintinib |
| | SAEs Leading to Dose Interruption of Fruquintinib |
| | SAEs Leading to Dose Interruption of Tislelizumab |
| | - SAEs Leading to Treatment Discontinuation of Fruquintinib |
| | SAEs Leading to Treatment Discontinuation of Tislelizumab |
| | - Fruquintinib -related SAEs Leading to Dose Reduction of Fruquintinib |
| | - Fruquintinib -related SAEs Leading to Dose Interruption of Fruquintinib |
| | Tislelizumab-related SAEs Leading to Dose Interruption of Tislelizumab |
| | - Fruquintinib-related SAEs Leading to Treatment Discontinuation of |
| | Fruquintinib |
| | - Tislelizumab-related SAEs Leading to Treatment Discontinuation of |
| | Tislelizumab |
| | - SAEs Leading to Death |
| Treatment- | <ul> <li>CTCAE Grade ≥3 AESIs</li> </ul> |
| emergent | - Fruquintinib-related AESIs |
| AESIs for | AESIs for Fruquintinib Leading to Dose Reduction of Fruquintinib |
| Fruquintinib | - AESIs for Fruquintinib Leading to Dose Interruption of Fruquintinib |
| | - AESIs for Fruquintinib Leading to Dose Interruption of Tislelizumab |
| | - AESIs for Fruquintinib Leading to Treatment Discontinuation of |
| | Fruquintinib |
| | - AESIs for Fruquintinib Leading to Treatment Discontinuation of |
| | Tislelizumab |
| | - Fruquintinib -related AESIs for Fruquintinib Leading to Dose Reduction |
| | of Fruquintinib |
| | Fruquintinib -related AESIs for Fruquintinib Leading to Dose |
| | Interruption of Fruquintinib |
| | Fruquintinib-related AESIs for Fruquintinib Leading to Treatment |
| | Discontinuation of Fruquintinib |
| | AESIs for Fruquintinib Leading to Death |
| Treatment- | <ul> <li>CTCAE Grade ≥3 imAEs</li> </ul> |
| related imAEs | imAEs for Tislelizumab Leading to Dose Reduction of Fruquintinib |
| to Tislelizumab | imAEs for Tislelizumab Leading to Dose Interruption of Fruquintinib |
| | imAEs for Tislelizumab Leading to Dose Interruption of Tislelizumab |
| | imAEs for Tislelizumab Leading to Treatment Discontinuation of |
| | Fruquintinib |
| | imAEs for Tislelizumab Leading to Treatment Discontinuation of |
| | Tislelizumab |
| | Tislelizumab-related imAEs for Tislelizumab Leading to Dose |
| | Interruption of Tislelizumab |

| Group | Summary scope |
|---|---|
| | - Tislelizumab-related imAEs for Tislelizumab Leading to Treatment |
| | Discontinuation of Tislelizumab |
| | - imAEs for Tislelizumab Leading to Death |
| COVID-19- | - CTCAE Grade ≥ 3 |
| related TEAEs | |

The number and percent of patients experiencing a TEAE within each of the categories and subcategories listed in Table above will be also summarized by SOC, PT, and highest CTCAE grade for each cohort. If a patient reports a TEAE more than once within that SOC/PT, the AE with the highest severity will be used in the corresponding severity summaries.

The summary will be sorted in descending order of frequency of SOC according to the sum of the column. Within the SOC, sorted by descending frequency of PT according to the sum of the column.

Time (days) to onset of the first treatment-emergent AESI will be descriptively summarized for each cohort.

All AEs, including AEs that started prior to the study drug, will be presented in patient listings. In addition, separate listings of all SAEs, AESIs, imAEs, AEs leading to death, drug-related AEs, AEs leading to dose reduction, AEs leading to dose interruption, and AEs leading to study drug discontinuation will be provided.

#### 5.2.11.3. Death

Number of deaths, primary cause of death and whether autopsy was performed are summarized descriptively for each cohort. Similarly, deaths which occur during the treatment period will also be tabulated.

Data for deaths will be provided as a patient list in which the on-treatment deaths will be flagged.

#### 5.2.11.4. Laboratory Evaluations

For hematology and clinical chemistry labs, the observed values and change from baseline will be summarized by visit using descriptive statistics.

Toxicities for clinical labs will be characterized according to CTCAE, v5.0 (Appendix 2), and the frequency and percentage of patients with each CTCAE grade for each visit during the treatment period will be described. Moreover, any occurrence of Grade 3 or Grade 4 during the overall treatment period will be summarized, and shift in grade from baseline to the worst post-baseline value will be summarized. Both the scheduled and unscheduled assessments will be used to identify the worst post-baseline values.

A summary table will be also provided for abnormal hepatic laboratory values by cohort. Abnormal hepatic laboratory values are based on the pre-specified thresholds (section 4.4.3).

Listings of all laboratory data with normal reference ranges, and CTCAE grades (when possible) will be provided.

 Date: 29 July 2024

#### 5.2.11.5. ECG

Descriptive statistics will be presented for each ECG parameter for the observed values and change from baseline to post baseline by visit.

A listing of all ECG data will be provided.

The criteria for potentially clinically significant findings are defined in Table 7. The frequency and percentage of patients with any potentially clinically significant findings during the treatment period will be presented. The supportive data will be provided in patient data listings.

#### 5.2.11.6. Vital Signs

For vital sign parameters (SBP, DBP, heart rate, temperature, and weight) the observed values and change from baseline will be summarized using descriptive statistics at each visit during the treatment period.

Additionally, the frequency and percentage of patients with any potentially clinically significant findings (defined in <u>Table 8</u>) during the overall treatment period will be presented. A listing of all vital sign data will be provided.

Moreover, the minimum, maximum, and their corresponding change from baseline vital sign values will be summarized descriptively overall treatment period.

#### 5.2.11.7. Performance Status

The frequency and percentage of patients for each ECOG score level will be summarized by visit. Shift in grade from baseline to the maximum post-baseline score will be summarized.

A listing of ECOG scores for all patients will be provided.

#### 5.2.11.8. Echocardiogram

Descriptive statistics for ECHO/MUGA will be summarized by visit. A by-patient listing of ECHO/MUGA values at each time point will be presented.

#### 5.2.11.9. Physical Examination

A listing of physical examination data for all patients will be provided.

#### 5.3. Subgroup Analyses

Not applicable.

#### 5.4. Other Analyses

#### 5.4.1. Pharmacokinetic Analysis

The PK analysis is used for listing and summaries of data specified in this section.

#### 5.4.1.1. Handling of Missing Data

Missing concentration data for all patients who are administered scheduled study treatments is considered as non-informative missing and will not be imputed. No concentration estimates will be provided for missing sample values.

#### 5.4.1.2. Handling of Dose Reduction or Interruption.

Any concentration data taken at or after the time of a dose reduced or interrupted of fruquintinib, or a dose interrupted of tislelizumab will be listed with a flag but excluded from summary statistics.

#### 5.4.1.3. Handling of below the lower limit of quantification (BLQ) Data

PK concentration summary, the following rules apply:

PK concentrations below the lower limit of quantification (BLQ) will be set to zero.

The following rules will apply for listing and presenting individual PK data:

- All concentrations are presented in original units and to the same decimal place as reported by Bioanalytical lab, e.g., ng/mL;
- Listing of PK sampling times including nominal and actual time elapsed from reference dose with the deviation from the nominal time and measured concentrations of the drug.
- If actual time is missing, time will be reported as NR (not recorded) and actual time will be reported as NC (not calculated). For fruquintinib, reference dose will be the fruquintinib dose on the day of fruquintinib PK sample collection. For tislelizumab, reference dose will be the tislelizumab dose during the same cycle of tislelizumab PK sample collection or last tislelizumab dose for EOT samples.

#### 5.4.1.4. Summary of PK concentration Data

Concentration data of fruquintinib, metabolite M11, and tislelizumab will be listed and summarized. Descriptive statistics will include number of patients [n], arithmetic mean, standard deviation, coefficient of variation [CV%], median, minimum, and maximum as appropriate.

The conventions presented in Table below are used for the presentation of the descriptive statistics of PK concentrations

| Variable | Summarized with: |
|---|---|
| Minimum, Maximum | 3 significant digits or as needed based on actual measured values |
| Mean (arithmetic), Median | 3 significant digits |
| StdDev | 3 significant digits |
| CV% | 1 decimal point |

# 5.4.1.5. Handling of the Difference between the Scheduled (nominal time) and the Actual Sampling Times (actual time)

For all sampling times, the actual sampling times relative to dosing will be calculated as the difference between the actual clock time of sampling and the actual clock time of dosing on the day of PK visit. For the visit when no dose administration is scheduled (e.g., no tislelizumab administration on C1D8 and C1D15), the actual sampling times will be calculated as the difference between the actual clock time of sampling and the actual clock time of the most recent dose administered prior to the visit (e.g., C1D1). If the actual time of sampling is missing, it will be reported as NR (not recorded) in the listing, the nominal time will be used for summary statistics.

#### 5.4.2. Immunogenicity Analysis

The Antidrug Antibody (ADA) analysis set are patients that have one baseline ADA measurement and at least one post-baseline ADA measurement.

The incidences of positive ADAs and neutralizing ADAs to tislelizumab will be reported for evaluable patients. When available, titer will be reported. The immunogenicity results will be summarized using descriptive statistics by the number and percentage of patients who develop detectable ADAs to tislelizumab according to the following attributes and endpoints.

#### ADA attributes:

- Treatment-boosted ADA is defined as ADA positive at baseline that was boosted to a 4fold or higher-level following drug administration.
- In order to calculate fold change, titer values reported as '<10' will be assigned a numerical value of 1.
- Treatment-induced ADA is defined as ADA negative at baseline and ADA positive post-baseline.
- Transient ADA response is defined as treatment-induced ADA detected only at 1 time point during treatment or follow-up, excluding last time point; or detected at 2 or more time points during treatment or follow-up, where the first and last positive samples are separated by less than 16 weeks and the last time point is negative.
- Persistent ADA response is defined as treatment-induced ADA detected at 2 or more time points during treatment or follow-up, where the first and last ADA positive samples are separated by 16 weeks or longer; or detected only in the last time point.
- Neutralizing ADA is defined as ADA that inhibits or reduces pharmacological activity.

#### ADA response endpoints:

- ADA incidence (also known as treatment-emergent ADA) is defined as sum of treatment-induced and treatment-boosted ADA-positive patients as a proportion of the ADA evaluable population.
- ADA prevalence is defined as proportion of all patients that are ADA positive, including pre-existing ADA, at any time point.

The following rules will apply for listing and presenting individual ADA data:

- All ADA results are presented as reported by the Bioanalytical lab, e.g., negative or
  positive and titer value (if applicable);
- Listing of ADA sampling times including nominal and actual time elapsed from
  tislelizumab dose with the deviation from the nominal time and ADA results by
  screening, confirmatory or titer (as applicable). If actual time is missing, time will be
  reported as NR (not recorded) and actual time will be reported as NC (not calculated).
  For ADA, reference dose will be the tislelizumab dose during the same cycle of ADA
  sample collection or last tislelizumab dose for EOT samples.

#### 5.4.3. Exploratory Analyses

Distribution of PD-L1 expression or MSS/MSI status will be examined in all patients. Other potential predictive markers including, but not limited to, TILs, TMB, cytokine expression, and gene signature profiling may be detected and analyzed.

Exploratory biomarker analyses will be performed in an effort to understand the association of these markers with study drug response, such as efficacy and resistance.

The biomarker data and analysis may be reported separately from the CSR.

#### 6. PLANNED ANALYSIS

#### 6.1. Independent Safety Data Monitoring

Safety monitoring and evaluation of the safety lead-in (Part 1) will be carried out by the Safety Review Committee (SRC). Safety will be evaluated to determine or confirm the RP2D for the combination of fruquintinib and tislelizumab.

After the RP2D has been determined in Part 1, the SRC will continue to periodically review the cumulative safety data during the conduct of Part 2.

#### 6.2. Interim Analysis

An interim analysis from Database Lock (DBL) was conducted to support the safety data review and regulatory interaction in the fruquintinib new drug application (NDA), the data snapshot was taken on column with data cutoff date on patients. By the time of the scheduled interim analysis, no patients were enrolled in the Part 2, therefore, the analysis was carried out only on patients from Part 1. Key study safety data collected up through the time of defined data cutoff were summarized.

#### 6.3. Final Analysis

The final analysis will be conducted after DBL for this study. All study data collected up through the time of the final analysis will be summarized, unless otherwise specified.

#### 7. CHANGE FROM THE PROTOCOL

A few noted changes from the protocol are summarized as follow:

- The pharmacokinetics analysis set definition has been updated compared to the protocol
  as some patients may have no fruquintinib samples as the appropriate blood collection
  tubes were not available. However, they will still have tislelizumab samples.
- Though in the protocol, it is stated that summary will only be conducted for these cohorts
  if there are more than 3 patients enrolled and dosed, in the actual table production, the
  summary information will still be presented for a cohort regardless of the number of
  patients enrolled for the cohort.
- The DLT- evaluable analysis set definition in the protocol is to include all patients enrolled into the safety lead-in portion of the study who meet at least one criteria of (i) and (ii), and both criteria (iii) and (iv) as defined as (i) received ≥85% of scheduled fruquintinib and ≥67% of scheduled tislelizumab administration during the DLT assessment window; (ii) experienced a DLT; (iii) did not receive prophylactic supportive care that confounds the evaluation of DLTs. That is, for a patient, if there is a record in concomitant medication with category being 'PRIOR AND CONCOMITANT MEDICATIONS', indication being 'PROPHYLAXIS', and the medication is taken within 28 days (≤ 28) since the date of first study drug administration, then the patient will be considered to have received preventive treatment during the DLT period; (iv) did not take a strong inducer of enzyme CYP3A. However, these criteria have been incorporated in the SRC review and it is aligned with those patients who took at one dose of study drug fruquintinib or tislelizumab. Therefore, the DLT-evaluable analysis set will be based on the decision from the SRC review and is defined to include all patients who took at one dose of study drug fruquintinib or tislelizumab.

#### REFERENCE

#### Allison 2020

Allison KH, Hammond EH, Dowsett M, et al. Estrogen and progesterone receptor testing in breast cancer: ASCO/CAP guideline update. J Clin Oncol. 2020;38:1346-66.

Brookmeyer 1982

Brookmeyer R., and Crowley J. (1982). A confidence interval for the median survival time. Biometrics, 29-41.

#### Eisenhauer 2009

Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumors: revised RECIST guideline (version 1.1). Eur J Cancer. 2009; 45:228-247.

#### Rakha 2014

Rakha EA, Starczynski J, Lee AHS, Ellis IO. The updated ASCO/CAP guideline recommendations for HER2 testing in the management of invasive breast cancer: a critical review of their implications for routine practice. Histopathology. 2014;64:609–615.

#### APPENDIX

#### Appendix 1: Study Schedule of Events

| Cycle/Period | | | | C | 1 | | | C2 | C3+ | ЕОТ | Safety<br>Follow-<br>up | Survival<br>Follow-<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Scre | ening | D1 | D8 | D15 | D21 | D1 | D15 | D1 | ≤7 Days<br>After<br>Last<br>Dose | 30 Days<br>After<br>EOT<br>Visit | Every<br>8 Weeks<br>After<br>EOT<br>Visit |
| Visit Window (days) | -28 to -1 | -7 to -1 | | ±1 | ±1 | ±1 | ±1 | ±1 | ±3 | ±3 | ±7 | ±14 |
| Informed consenta | X | | | | | | | | | | | |
| PD-L1 expression<br>confirmation <sup>b</sup> | X | | | | | | | | | | | |
| MSS/MSI status<br>confirmation <sup>c</sup> | X | | | | | | | | | | | |
| Medical history, disease<br>history <sup>d</sup> | х | | | | | | | | | | | |
| Demographicse | X | | | | | | | | | | | |
| Prior and concomitant<br>medications and<br>concomitant procedures <sup>f</sup> | X | | X | X | X | X | X | X | X | X | X | |
| Comprehensive physical examination <sup>g</sup> | X | | X | | | | | | | | | |
| Limited physical examination <sup>h</sup> | | | | X | X | X | X | | X | X | X | |
| Vital signs <sup>i</sup> | X | | X | X | X | х | х | x | X | x | X | |
| ECOG performance statusi | | X | X | | | | X | | X | X | X | |
| Laboratory evaluations: | | X | | | | | | | | | | |
| Hematology <sup>j</sup> | | X | | X | X | X | X | X | X | X | | |
| Blood chemistryk | | X | | X | X | X | X | X | X | X | | |

| Cycle/Period | | | | C | 1 | | • | C2 | C3+ | ЕОТ | Safety<br>Follow-<br>up | Survival<br>Follow-<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Scre | ening | D1 | D8 | D15 | D21 | D1 | D15 | D1 | ≤7 Days<br>After<br>Last<br>Dose | 30 Days<br>After<br>EOT<br>Visit | Every<br>8 Weeks<br>After<br>EOT<br>Visit |
| Visit Window (days) | -28 to -1 | -7 to -1 | | ±1 | ±1 | ±1 | ±1 | ±1 | ±3 | ±3 | ±7 | ±14 |
| Blood amylase and<br>lipase | | X | | X | X | | х | X | X | х | | |
| Fasting lipid panel <sup>l</sup> | | X | | | | | X | | X | X | | |
| Coagulation indicators <sup>m</sup> | | X | | X | X | X | X | X | X | X | | |
| Serum pregnancy test <sup>n</sup> | | X | | | | | | | | | X | |
| Urine pregnancy test <sup>n</sup> | | | X | | | | X | | X | X | | |
| Thyroid function test <sup>o</sup> | X | | | | X | | X | X | X | | | |
| Urinalysis <sup>p</sup> | | X | | | | X | X | | X | | | |
| Virological screening <sup>q</sup> | X | | | | | | | | X | X | | |
| PK assessments | | | | | | Refer | to protocol | Table 2 | | | | |
| Tislelizumab<br>immunogenicity | | | | | | Refer | to protocol | Table 2 | | | | |
| 12-Lead ECG <sup>r</sup> | X | | | | X | | X | | X | | X | |
| ECHO/MUGA scan | X | | | Every 12 | weeks from | C1D1 (±1 v | week) until | progression o | of disease | | | |
| Tumor evaluation/imaging <sup>5</sup> | | Screening | ng and every | 8 weeks (±1 | l week) from | C1D1 until | disease pro | gression | | X | | |
| Fruquintinib drug<br>administration | | | | PO QD, Days 1 to 21 of each cycle | | | | | | | | |
| Tislelizumab drug<br>administration <sup>†</sup> | | | Х | | | | X | | Х | | | |
| AEs/SAEs <sup>u</sup> | X | | X | X | X | X | X | X | X | X | X | |
| Overall survival <sup>v</sup> | | | | | | | | | | | | X |

Study Protocol: 2020-013-00US3

AE=adverse event, ALP=alkaline phosphatase; ALT=alanine aminotransferase; aPTT=activated partial thromboplastin time; AST=aspartate aminotransferase; C=cycle; CK=creatine kinase; CKMB=creatine kinase-MB; CrCl=creatinine clearance; D=day; DNA=deoxyribonucleic acid; ECG=electrocardiogram; ECHO=echocardiogram; ECGG=eastern cooperative oncology group; eCRF=electronic case report form; EOT=end of treatment; HBV=hepatitis B virus; HBsAg=hepatitis B surface antigen; HCV=hepatitis C virus; HIV=human immunodeficiency virus; ICF=informed consent form; INR=international normalized ratio; IV=intravenous; MSI=microsatellite instability; MSS=microsatellite stability stable; MUGA=multigated acquisition; PCR=polymerase chain reaction; PD=progressive disease; PD-L1=programmed death-ligand 1; PK=pharmacokinetics; PO=orally; QD=once daily; Q3W=every 3 weeks; Q4W=every 4 weeks; QTcF=QT interval corrected by the method of Fredericia; RNA=ribonucleic acid; RP2D=recommended phase 2 dose; SAE=serious adverse event; SOP=standard operating procedure.

- Written informed consent must be obtained before any study-related examinations or procedures are performed. However, before informed consent is obtained, if the examinations for standard treatment are performed within 28 days before the planned C1D1, they can be used to replace the examinations during the screening period without repeating the examinations, except for examinations that need to be performed 7 days before the start of the study drug administration.
- b PD-L1 expression as determined locally, for Cohorts A, B, and C. The results should be available in the source documents and be those used to make treatment decisions for the patient. A redacted copy of the local results should accompany the archival tumor samples submitted as part of the protocol.
- MSS/MSI status as determined locally, for Cohorts C and D only. The results should be available in the source documents and be those used to make treatment decisions for the patient. A redacted copy of the local results should accompany the archival tumor samples submitted as part of the protocol.
- Medical history and disease history data include significant clinical disease or symptom, surgical history, history of malignancy (including date of diagnosis, classification and prognosis evaluation of the study disease, and the treatment performed and the outcome; the tumor species and outcomes of any other previous malignancies), smoking history, history of alcohol consumption, history of drug abuse, and other medical-related history.
- Demographic information includes sex, race, and in some countries, year of birth.
- Concomitant medications include any prescription and over-the-counter medications started after signing of ICF. During the screening period, all drugs used for the patient within 28 days prior to the start of study drug should be recorded. In subsequent visits, the drugs used in the patient after the last record, as well as drugs 30 days after the last dose of study drug(s), should be recorded in eCRF. Subsequent new anti-tumor treatment regimens during the Safety and Survival Follow-up Periods will also be recorded.
- A comprehensive physical examination includes patient height, weight, and general condition, as well as an examination of the head, heart, chest (including the lungs), abdomen, extremities, skin, lymph nodes, nervous system, and additional areas/systems as clinically indicated.
- Limited physical examination includes vital signs and any change from baseline; any new abnormalities; examination of weight, thorax, abdomen; and additional areas/systems as clinically indicated. In order to assess changes from baseline and to evaluate for new abnormalities, the limited physical examination should assess for new or changed skin lesions, enlarged lymph nodes, palpable masses, and appropriate examination to address any patient-reported symptoms.
- Assessments can be performed up to and including C1D1. Details for ECOG assessment can be found in Section 6.1.11 of the protocol and for vital sign collection in Section 6.1.12 of the protocol.
- Hematology includes red blood cell count, hemoglobin, hematocrit, absolute reticulocyte count, white blood cell count and classifications (neutrophils, lymphocytes, eosinophils, monocytes, and basophils), and platelet count. If abnormal or primitive immature cells are seen, they must also be recorded. Any additional routine blood tests during the study shall be arranged by the investigator as needed.
- Blood chemistry includes ALT, AST, alkaline phosphatase (ALP), bicarbonate, bilirubin/total bilirubin, lactic dehydrogenase, non-fasting total cholesterol, triglycerides, uric acid, total protein, albumin, blood urea nitrogen or urea, creatinine, CrCl rate, sodium, potassium, magnesium, chloride, corrected calcium (for patients with hypoproteinemia), phosphorus, blood glucose, creatine phosphokinase, and creatine kinase-MB (CK-MB). If CK-MB fractionation is not available, troponin I and/or troponin T should be tested instead. Serum troponins may be substituted per local guidelines if used consistently throughout the study. If tislelizumab has been permanently discontinued, CK and CK-MB testing will be done as clinically indicated.
- Fasting lipid panel includes total cholesterol, high-density lipoprotein, low-density lipoprotein, and triglycerides.
- <sup>m</sup> Coagulation indicators include prothrombin time, aPTT, and INR.
- Female patients of childbearing potential (including those who have undergone tubal ligation) must undergo a serum pregnancy test ≤7 days before the first dose and record a negative result. If serum pregnancy test was drawn within 72 hours of C1D1, then urine pregnancy test is not required on C1D1. After enrollment, urine pregnancy test should be conducted on Day 1 of every treatment cycle starting from Cycle 1, and at the EOT visit. A serum pregnancy test should be performed at the Safety Follow-up Visit. If the result of urine pregnancy testing is equivocal, a serum test should be performed. Unscheduled testing via either method can be performed if there is an indication, however, any equivocal urine pregnancy tests should be repeated via serum pregnancy testing.

- Thyroid function tests include serum free tri-iodothyronine, serum free thyroxine, and thyroid stimulating hormone.
- P Urinalysis includes urine pH, protein, glucose, blood and ketones; microscopic for white blood cell and red blood cell count. A 24-hour urine for quantitative protein must be collected from all patients with 1+ proteinuria.
- Testing will be performed by the local laboratory at screening and will include HBV/HCV serology (HBsAg and HCV antibody) and viral load assessment (HBV DNA and HCV RNA), which will be assessed only when HBsAg or HCV antibody is positive, respectively. Additionally, for patients who have detectable HBV DNA at screening, the respective viral load test will be performed every 4 cycles starting at Cycle 5 (ie, Day 1 of Cycles 5, 9, 13, etc) and at the EOT visit.
- ECG indicators include PR interval, QRS interval, RR interval, QT/QTcF interval and heart rate. Unscheduled ECG or other cardiac examinations can be performed if clinically indicated. All ECGs should be done prior to dosing of study drugs.
- If a patient discontinues study drug(s) due to reasons other than PD or death, tumor assessments should continue to be performed following the scheduled assessment plan until the start of new anticancer therapy, PD, death, lost to follow-up, or withdrawal of consent...
- Tislelizumab 300 mg IV will be administered on Day 1 of each 28-day cycle (once every 4 weeks). Every 3 weeks (Q3W) dosing of tislelizumab may be explored depending on the tolerability of the Q4W dosing schedule.
- After signing the informed consent form, all AEs including SAEs regardless of attribution will be collected until 30 days after the last dose of study drug or initiation of a new treatment therapy, whichever is earlier. After this period, investigators should report only SAEs that are considered to be related to the study drug. Immune-mediated AEs (serious or nonserious) should be reported until 90 days after the last dose of tislelizumab regardless of whether or not the patient starts a new anticancer therapy.
- Following EOT, patients will be followed every 8 weeks (±14 days) via telephone or in manner that follows local site SOPs.

Appendix 2: CTCAE criteria table for lab parameters

| | | | | ATOXGI | ATOXGR | |
|---|---|---|---|---|---|---|
| PARAM (SI Unit) | Нуро | Hyper | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
| | | Hemoglobin increased | Increase in >0 - 2 g/dL | Increase in >2 - 4<br>g/dL | Increase in >4 g/dL | ~ |
| Hemoglobin (g/L) | Anemia | | Hemoglobin (Hgb) <lln -="" 10.0="" 100="" 6.2="" <lln="" dl;="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0<br/>g/dL;<br/>&lt;6.2 - 4.9 mmol/L;<br/>&lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL;<br/>&lt;4.9 mmol/L;<br/>&lt;80 g/L</td><td>~</td></lln> | Hgb <10.0 - 8.0<br>g/dL;<br><6.2 - 4.9 mmol/L;<br><100 - 80g/L | Hgb <8.0 g/dL;<br><4.9 mmol/L;<br><80 g/L | ~ |
| Platelets (10^9/L) | Platelet count<br>decreased | | <lln -="" 75,000="" mm3;<br=""><lln -="" 10e9="" 75.0="" l<="" td="" x=""><td>&lt;75,000 -<br/>50,000/mm3; &lt;75.0 -<br/>50.0 x 10e9 /L</td><td>&lt;50,000 -<br/>25,000/mm3; &lt;50.0<br/>- 25.0 x 10e9 /L</td><td>&lt;25,000/mm3;<br/>&lt;25.0 x 10e9 /L</td></lln></lln> | <75,000 -<br>50,000/mm3; <75.0 -<br>50.0 x 10e9 /L | <50,000 -<br>25,000/mm3; <50.0<br>- 25.0 x 10e9 /L | <25,000/mm3;<br><25.0 x 10e9 /L |
| Leukocytes (10^9/L) | White blood cell<br>decreased | | <lln -="" 3000="" mm3;<br=""><lln -="" 10e9="" 3.0="" l<="" td="" x=""><td>&lt;3000 - 2000/mm3;<br/>&lt;3.0 - 2.0 x 10e9 /L</td><td>&lt;2000 - 1000/mm3;<br/>&lt;2.0 - 1.0 x 10e9 /L</td><td>&lt;1000/mm3;<br/>&lt;1.0 x 10e9 /L</td></lln></lln> | <3000 - 2000/mm3;<br><3.0 - 2.0 x 10e9 /L | <2000 - 1000/mm3;<br><2.0 - 1.0 x 10e9 /L | <1000/mm3;<br><1.0 x 10e9 /L |
| Neutrophils (10^9/L) | Neutrophil count<br>decreased | | <lln -="" 1500="" mm3;<br=""><lln -="" 1.5="" 10e9="" l<="" td="" x=""><td>&lt;1500 - 1000/mm3;<br/>&lt;1.5 - 1.0 x 10e9 /L</td><td>&lt;1000 - 500/mm3;<br/>&lt;1.0 - 0.5 x 10e9 /L</td><td>&lt;500/mm3;<br/>&lt;0.5 x 10e9 /L</td></lln></lln> | <1500 - 1000/mm3;<br><1.5 - 1.0 x 10e9 /L | <1000 - 500/mm3;<br><1.0 - 0.5 x 10e9 /L | <500/mm3;<br><0.5 x 10e9 /L |
| Lymphocytes | Lymphocyte count decreased | | <lln -="" 800="" mm3;<br=""><lln -="" 0.8="" 10e9="" l<="" td="" x=""><td>&lt;800 - 500/mm3;<br/>&lt;0.8 - 0.5 x 10e9 /L</td><td>&lt;500 - 200/mm3;<br/>&lt;0.5 - 0.2 x 10e9 /L</td><td>&lt;200/mm3;<br/>&lt;0.2 x 10e9 /L</td></lln></lln> | <800 - 500/mm3;<br><0.8 - 0.5 x 10e9 /L | <500 - 200/mm3;<br><0.5 - 0.2 x 10e9 /L | <200/mm3;<br><0.2 x 10e9 /L |
| (10^9/L) | | Lymphocyte count increased | ~ | >4000/mm3 -<br>20,000/mm3 | >20,000/mm3 | ~ |
| Eosinophils (%) | | Eosinophilia | >ULN and >Baseline | - | Steroids initiated | - |
| Activated Partial<br>Thromboplastin Time<br>(s) | | Activated partial thromboplastin time prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN;<br>bleeding | ~ |
| International<br>Normalized Ratio | | INR increased | >1.2 - 1.5 | >1.5 - 2.5 | >2.5 | ~ |
| Albumin (g/L) | Hypoalbuminemia | | <lln -="" -<br="" 3="" <lln="" dl;="" g="">30 g/L</lln> | <3 - 2 g/dL; <30 - 20<br>g/L | <2 g/dL; <20 g/L | ~ |
| Glucose (mmol/L) | Hypoglycemia | | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 - 40 mg/dL;<br/>&lt;3.0 - 2.2 mmol/L</td><td>&lt;40 - 30 mg/dL;<br/>&lt;2.2 - 1.7 mmol/L</td><td>&lt;30 mg/dL;<br/>&lt;1.7 mmol/L</td></lln></lln> | <55 - 40 mg/dL;<br><3.0 - 2.2 mmol/L | <40 - 30 mg/dL;<br><2.2 - 1.7 mmol/L | <30 mg/dL;<br><1.7 mmol/L |

| | | | | ATOXGI | ₹ | |
|---|---|---|---|---|---|---|
| PARAM (SI Unit) | Нуро | Hyper | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
| Creatinine (umol/L) | | Creatinine increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x baseline<br>if baseline was<br>abnormal; >1.5 - 3.0<br>x ULN if baseline<br>was normal | >3.0 x baseline-<br>6.0xULN if baseline<br>was abnormal; >3.0<br>- 6.0 x ULN if<br>baseline is normal | >6.0 x ULN |
| Creatine<br>phosphokinase (IU/L) | | CPK increased | >ULN - 2.5 x ULN | >2.5 x ULN- 5 x<br>ULN | >5.0 X ULN - 10.0<br>x ULN | >10.0 x ULN |
| Alkaline Phosphatase<br>(uKat/L) | | Alkaline phosphatase increased | >ULN - 2.5 x ULN if<br>baseline was normal;<br>2.0 - 2.5 x baseline if<br>baseline was abnormal | >2.5 - 5.0 x ULN if<br>baseline was normal;<br>>2.5 - 5.0 x baseline<br>if baseline was<br>abnormal | >5.0 - 20.0 x ULN<br>if baseline was<br>normal; >5.0 - 20.0<br>x baseline if<br>baseline was<br>abnormal | >20.0 x ULN if<br>baseline was<br>normal; >20.0 x<br>baseline if<br>baseline was<br>abnormal |
| Aspartate<br>Aminotransferase<br>(uKat/L) | | Aspartate<br>aminotransferase<br>increased | >ULN - 3.0 x ULN if<br>baseline was normal;<br>1.5 - 3.0 x baseline if<br>baseline was abnormal | >3.0 - 5.0 x ULN if<br>baseline was normal;<br>>3.0 - 5.0 x baseline<br>if baseline was<br>abnormal | >5.0 - 20.0 x ULN<br>if baseline was<br>normal; >5.0 - 20.0<br>x baseline if<br>baseline was<br>abnormal | >20.0 x ULN if<br>baseline was<br>normal; >20.0 x<br>baseline if<br>baseline was<br>abnormal |
| Alanine<br>Aminotransferase<br>(uKat/L) | | Alanine<br>aminotransferase<br>increased | >ULN - 3.0 x ULN if<br>baseline was normal;<br>1.5 - 3.0 x baseline if<br>baseline was abnormal | >3.0 - 5.0 x ULN if<br>baseline was normal;<br>>3.0 - 5.0 x baseline<br>if baseline was<br>abnormal | >5.0 - 20.0 x ULN<br>if baseline was<br>normal; >5.0 - 20.0<br>x baseline if<br>baseline was<br>abnormal | >20.0 x ULN if<br>baseline was<br>normal; >20.0 x<br>baseline if<br>baseline was<br>abnormal |
| Serum Calcium | | Hypercalcemia | >ULN - 2.9 mmol/L | >2.9 - 3.1 mmol/L | >3.1 - 3.4 mmol/L | >3.4 mmol/L |
| (mmol/L) | Hypocalcemia | | <lln -="" 2.0="" l<="" mmol="" td=""><td>&lt;2.0 - 1.75 mmol/L</td><td>&lt;1.75 - 1.5 mmol/L</td><td>&lt;1.5 mmol/L</td></lln> | <2.0 - 1.75 mmol/L | <1.75 - 1.5 mmol/L | <1.5 mmol/L |
| Magnesium | | Hypermagnesemia | >ULN - 3.0 mg/dL;<br>>ULN - 1.23 mmol/L | ~ | >3.0 - 8.0 mg/dL;<br>>1.23 - 3.30<br>mmol/L | >8.0 mg/dL;<br>>3.30 mmol/L |
| (mmol/L) | Hypomagnesemia | | <lln -="" 1.2="" dl;<br="" mg=""><lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL;<br/>&lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 - 0.7 mg/dL;<br/>&lt;0.4 - 0.3 mmol/L</td><td>&lt;0.7 mg/dL;<br/>&lt;0.3 mmol/L</td></lln></lln> | <1.2 - 0.9 mg/dL;<br><0.5 - 0.4 mmol/L | <0.9 - 0.7 mg/dL;<br><0.4 - 0.3 mmol/L | <0.7 mg/dL;<br><0.3 mmol/L |
| Potassium (mmol/L) | | Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L | >7.0 mmol/L |
| rotassium (mmort) | Hypokalemia | | <lln -="" 3.0="" l<="" mmol="" td=""><td>~</td><td>&lt;3.0 - 2.5 mmol/L</td><td>&lt;2.5 mmol/L</td></lln> | ~ | <3.0 - 2.5 mmol/L | <2.5 mmol/L |

| | | | | ATOXGI | 2 | |
|---|---|---|---|---|---|---|
| PARAM (SI Unit) | Нуро | Hyper | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
| S = 1: (1/T.) | | Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L | >160 mmol/L |
| Sodium (mmol/L) | Hyponatremia | | <lln -="" 130="" l<="" mmol="" td=""><td>125-129 mmol/L</td><td>120-124 mmol/L</td><td>&lt;120 mmol/L</td></lln> | 125-129 mmol/L | 120-124 mmol/L | <120 mmol/L |
| Total cholesterol<br>(mmol/L) | | Cholesterol high | >ULN - 300 mg/dL;<br>>ULN - 7.75 mmol/L | >300 - 400 mg/dL;<br>>7.75 - 10.34<br>mmol/L | >400 - 500 mg/dL;<br>>10.34 - 12.92<br>mmol/L | >500 mg/dL;<br>>12.92 mmol/L |
| Bilirubin (umol/L) | | Blood bilirubin increased | >ULN - 1.5 x ULN if<br>baseline was normal; ><br>1.0 - 1.5 x baseline if<br>baseline was abnormal | >1.5 - 3.0 x ULN if<br>baseline was normal;<br>>1.5 - 3.0 x baseline<br>if baseline was<br>abnormal | >3.0 - 10.0 x ULN<br>if baseline was<br>normal; >3.0 - 10.0<br>x baseline if<br>baseline was<br>abnormal | >10.0 x ULN if<br>baseline was<br>normal; >10.0 x<br>baseline if<br>baseline was<br>abnormal |
| Triglycerides<br>(mmol/L) | | Hypertriglyceridemia | 150 mg/dL - 300<br>mg/dL; 1.71 mmol/L -<br>3.42 mmol/L | >300 mg/dL - 500<br>mg/dL; >3.42<br>mmol/L - 5.7<br>mmol/L | >500 mg/dL - 1000<br>mg/dL; >5.7<br>mmol/L - 11.4<br>mmol/L | >1000 mg/dL;<br>>11.4 mmol/L |
| Urinary protein | | Proteinuria | 1+ proteinuria; urinary<br>protein ≥ULN - <1.0<br>g/24 hrs | 2+ and 3+<br>proteinuria; urinary<br>protein 1.0-<br><3.5g/24hrs | 4+ proteinuria;<br>urinary protein >=<br>3.5g/24hrs | ~ |

## Appendix 3: MedDRA (Version 25.0) Preferred Term List for AESI Categories

| | AESI Category: Thyroid Dysfunction | |
|---|---|---|
| Anti-thyroid antibody | Malignant exophthalmos | Thyroid stimulating hormone deficiency |
| Anti-thyroid antibody decreased | Marine Lenhart syndrome | Thyroid stimulating immunoglobulin increased |
| Anti-thyroid antibody increased | Multifocal fibrosclerosis | Thyroid therapy |
| Anti-thyroid antibody positive | Myxoedema | Thyroid tuberculosis |
| Antithyroid arthritis syndrome | Myxoedema coma | Thyroidectomy |
| Atrophic thyroiditis | Orbital decompression | Thyroiditis |
| Autoimmune hypothyroidism | Photon radiation therapy to thyroid | Thyroiditis acute |
| Autoimmune thyroid disorder | Polyglandular autoimmune syndrome type II | Thyroiditis chronic |
| Autoimmune thyroiditis | Polyglandular autoimmune syndrome type III | Thyroiditis fibrous chronic |
| Basedow's disease | Post procedural hypothyroidism | Thyroiditis subacute |
| Biopsy thyroid gland abnormal | Primary hyperthyroidism | Thyrotoxic cardiomyopathy |
| Blood thyroid stimulating hormone abnormal | Primary hypothyroidism | Thyrotoxic crisis |
| Blood thyroid stimulating hormone decreased | Protein bound iodine decreased | Thyrotoxic myopathy |
| Blood thyroid stimulating hormone increased | Protein bound iodine increased | Thyrotoxic periodic paralysis |
| Butanol-extractable iodine decreased | Radioactive iodine therapy | Thyroxin binding globulin abnormal |
| Butanol-extractable iodine increased | Radiotherapy to thyroid | Thyroxin binding globulin decreased |
| Central hypothyroidism | Reverse tri-iodothyronine decreased | Thyroxin binding globulin increased |
| Congenital hypothyroidism | Reverse tri-iodothyronine increased | Thyroxine abnormal |
| Congenital thyroid disorder | Secondary hyperthyroidism | Thyroxine decreased |
| Endocrine ophthalmopathy | Silent thyroiditis | Thyroxine free abnormal |
| Euthyroid sick syndrome | Thyreostatic therapy | Thyroxine free decreased |
| Exophthalmos | Thyroglobulin absent | Thyroxine free increased |
| Free thyroxine index abnormal | Thyroglobulin decreased | Thyroxine increased |
| Free thyroxine index decreased | Thyroglobulin increased | Thyroxine therapy |
| Free thyroxine index increased | Thyroglobulin present | Toxic goitre |
| Gamma radiation therapy to thyroid | Thyroid atrophy | Toxic nodular goitre |
| Generalised resistance to thyroid hormone | Thyroid autotransplantation | Transient hypothyroxinaemia of prematurity |
| Goitre | Thyroid dermatopathy | Tri-iodothyronine abnormal |
| Hashimoto's encephalopathy | Thyroid disorder | Tri-iodothyronine decreased |
| Hashitoxicosis | Thyroid dysfunction in pregnancy | Tri-iodothyronine free abnormal |
| Hyperthyroidism | Thyroid electron radiation therapy | Tri-iodothyronine free decreased |
| Hypothyroidic goitre | Thyroid function test abnormal | Tri-iodothyronine free increased |
| Hypothyroidism | Thyroid gland scan abnormal | Tri-iodothyronine free normal |
| Immune-mediated hyperthyroidism | Thyroid hemiagenesis | Tri-iodothyronine increased |
| Immune-mediated hypothyroidism | Thyroid hormone replacement therapy | Tri-iodothyronine uptake abnormal |

| Immune-mediated thyroiditis | Thyroid hormones decreased | Tri-iodothyronine uptake decreased |
|---|---|---|
| Inappropriate thyroid stimulating hormone secretion | Thyroid hormones increased | Tri-iodothyronine uptake increased |
| Infectious thyroiditis | Thyroid operation | Ultrasound thyroid abnormal |
| Iodine uptake abnormal | Thyroid pain | X-ray therapy to thyroid |
| Iodine uptake decreased | Thyroid releasing hormone challenge test abnormal | |
| Iodine uptake increased | Thyroid size decreased | |
| | _ | |
| | AESI Category: Proteinuria | |
| Albumin globulin ratio increased | Beta 2 microglobulin urine increased | Protein urine |
| Albumin urine present | Globulinuria | Protein urine present |
| Albuminuria | Microalbuminuria | Proteinuria |
| Bence Jones protein urine present | Myoglobinuria | Urine albumin/creatinine ratio increased |
| Bence Jones proteinuria | Orthostatic proteinuria | Urine protein/creatinine ratio abnormal |
| | | Urine protein/creatinine ratio increased |
| | AESI Category: Hypertension | |
| Accelerated hypertension | Hypertension neonatal | Metabolic syndrome |
| Blood pressure ambulatory increased | Hypertensive angiopathy | Neurogenic hypertension |
| Blood pressure diastolic increased | Hypertensive cardiomegaly | Orthostatic hypertension |
| Blood pressure inadequately controlled | Hypertensive cardiomyopathy | Page kidney |
| Blood pressure increased | Hypertensive cerebrovascular disease | Postoperative hypertension |
| Blood pressure management | Hypertensive crisis | Pre-eclampsia |
| Blood pressure orthostatic increased | Hypertensive emergency | Prehypertension |
| Blood pressure systolic increased | Hypertensive encephalopathy | Procedural hypertension |
| Catecholamine crisis | Hypertensive end-organ damage | Renal hypertension |
| Dialysis induced hypertension | Hypertensive heart disease | Renal sympathetic nerve ablation |
| Diastolic hypertension | Hypertensive nephropathy | Renovascular hypertension |
| Eclampsia | Hypertensive urgency | Retinopathy hypertensive |
| Endocrine hypertension | Labile hypertension | Secondary aldosteronism |
| Essential hypertension | Malignant hypertension | Secondary hypertension |
| Gestational hypertension | Malignant hypertensive heart disease | Superimposed pre-eclampsia |
| HELLP syndrome | Malignant renal hypertension | Supine hypertension |
| Hyperaldosteronism | Maternal hypertension affecting foetus | Systolic hypertension |
| Hypertension | Mean arterial pressure increased | Withdrawal hypertension |
| | AESI Category: Haemorrhages | |
| Abdominal wall haematoma | Haemophilic pseudotumour | Peritoneal haematoma |
| Abdominal wall haemorrhage | Haemoptysis | Periventricular haemorrhage neonatal |

| Abnormal uterine bleeding | Haemorrhage | Petechiae |
|---|---|---|
| Abnormal withdrawal bleeding | Haemorrhage coronary artery | Pharyngeal contusion |
| Achenbach syndrome | Haemorrhage foetal | Pharyngeal haematoma |
| Acute haemorrhagic leukoencephalitis | Haemorrhage in pregnancy | Pharyngeal haemorrhage |
| Acute haemorrhagic ulcerative colitis | Haemorrhage intracranial | Pituitary apoplexy |
| Administration site bruise | Haemorrhage neonatal | Pituitary haemorrhage |
| Administration site haematoma | Haemorrhage subcutaneous | Placenta praevia haemorrhage |
| Administration site haemorrhage | Haemorrhage subepidermal | Plasmin increased |
| Adrenal haematoma | Haemorrhage urinary tract | Polymenorrhagia |
| Adrenal haemorrhage | Haemorrhagic adrenal infarction | Post abortion haemorrhage |
| Anal fissure haemorrhage | Haemorrhagic arteriovenous malformation | Post procedural contusion |
| Anal haemorrhage | Haemorrhagic ascites | Post procedural haematoma |
| Anal ulcer haemorrhage | Haemorrhagic breast cyst | Post procedural haematuria |
| Anastomotic haemorrhage | Haemorrhagic cerebellar infarction | Post procedural haemorrhage |
| Anastomotic ulcer haemorrhage | Haemorrhagic cerebral infarction | Post transfusion purpura |
| | _ | Post-traumatic punctate intraepidermal |
| Aneurysm ruptured | Haemorrhagic cyst | haemorrhage |
| Angina bullosa haemorrhagica | Haemorrhagic diathesis | Postmenopausal haemorrhage |
| Anorectal varices haemorrhage | Haemorrhagic disease of newborn | Postpartum haemorrhage |
| Anticoagulant-related nephropathy | Haemorrhagic disorder | Prekallikrein increased |
| Antiplatelet reversal therapy | Haemorrhagic erosive gastritis | Premature separation of placenta |
| Aortic aneurysm rupture | Haemorrhagic gastroenteritis | Procedural haemorrhage |
| Aortic dissection rupture | Haemorrhagic hepatic cyst | Proctitis haemorrhagic |
| Aortic intramural haematoma | Haemorrhagic infarction | Prostatic haemorrhage |
| Aortic perforation | Haemorrhagic necrotic pancreatitis | Pulmonary alveolar haemorrhage |
| Aortic rupture | Haemorrhagic occlusive retinal vasculitis | Pulmonary contusion |
| Aponeurosis contusion | Haemorrhagic ovarian cyst | Pulmonary haematoma |
| Application site bruise | Haemorrhagic stroke | Pulmonary haemorrhage |
| Application site haematoma | Haemorrhagic thyroid cyst | Pulmonary haemorrhage neonatal |
| Application site haemorrhage | Haemorrhagic transformation stroke | Puncture site bruise |
| Application site purpura | Haemorrhagic tumour necrosis | Puncture site haematoma |
| Arterial haemorrhage | Haemorrhagic urticaria | Puncture site haemorrhage |
| Arterial intramural haematoma | Haemorrhagic vasculitis | Purpura |
| Arterial perforation | Haemorrhoidal haemorrhage | Purpura fulminans |
| Arterial rupture | Haemostasis | Purpura neonatal |
| Arteriovenous fistula site haematoma | Haemothorax | Purpura non-thrombocytopenic |
| Arteriovenous fistula site haemorrhage | Heavy menstrual bleeding | Purpura senile |
| Arteriovenous graft site haematoma | Henoch-Schonlein purpura | Putamen haemorrhage |

| Arteriovenous graft site haemorrhage | Hepatic artery haemorrhage | Radiation associated haemorrhage |
|---|---|---|
| Astringent therapy | Hepatic haemangioma rupture | Rectal haemorrhage |
| Atrial rupture | Hepatic haematoma | Rectal ulcer haemorrhage |
| Auricular haematoma | Hepatic haemorrhage | Renal artery perforation |
| Basal ganglia haematoma | Hereditary haemorrhagic telangiectasia | Renal cyst haemorrhage |
| Basal ganglia haemorrhage | Hyperfibrinolysis | Renal haematoma |
| | Hypergammaglobulinaemic purpura of | |
| Basilar artery perforation | Waldenstrom | Renal haemorrhage |
| Bladder tamponade | Hyphaema | Respiratory tract haemorrhage |
| Bleeding varicose vein | Iliac artery perforation | Respiratory tract haemorrhage neonatal |
| Blood blister | Iliac artery rupture | Retinal aneurysm rupture |
| Blood loss anaemia | Iliac vein perforation | Retinal haemorrhage |
| Blood urine | Immune thrombocytopenia | Retinopathy haemorrhagic |
| Blood urine present | Implant site bruising | Retroperitoneal haematoma |
| Bloody discharge | Implant site haematoma | Retroperitoneal haemorrhage |
| Bloody peritoneal effluent | Implant site haemorrhage | Retroplacental haematoma |
| Bone contusion | Incision site haematoma | Ruptured cerebral aneurysm |
| Bone marrow haemorrhage | Incision site haemorrhage | Scleral haematoma |
| Brain contusion | Increased tendency to bruise | Scleral haemorrhage |
| Brain stem haematoma | Induced abortion haemorrhage | Scrotal haematocoele |
| Brain stem haemorrhage | Inferior vena cava perforation | Scrotal haematoma |
| Brain stem microhaemorrhage | Infusion site bruising | Scrotal haemorrhage |
| Breast haematoma | Infusion site haematoma | Shock haemorrhagic |
| Breast haemorrhage | Infusion site haemorrhage | Skin haemorrhage |
| Broad ligament haematoma | Injection site bruising | Skin neoplasm bleeding |
| Bronchial haemorrhage | Injection site haematoma | Skin ulcer haemorrhage |
| Bronchial varices haemorrhage | Injection site haemorrhage | Small intestinal haemorrhage |
| Bullous haemorrhagic dermatosis | Instillation site bruise | Small intestinal ulcer haemorrhage |
| Bursal haematoma | Instillation site haematoma | Soft tissue haemorrhage |
| Cardiac contusion | Instillation site haemorrhage | Spermatic cord haemorrhage |
| Carotid aneurysm rupture | Intermenstrual bleeding | Spinal cord haematoma |
| Carotid artery perforation | Internal haemorrhage | Spinal cord haemorrhage |
| Catheter site bruise | Intestinal haematoma | Spinal epidural haematoma |
| Catheter site haematoma | Intestinal haemorrhage | Spinal epidural haemorrhage |
| Catheter site haemorrhage | Intestinal varices haemorrhage | Spinal subarachnoid haemorrhage |
| Central nervous system haemorrhage | Intra-abdominal haematoma | Spinal subdural haematoma |
| Cephalhaematoma | Intra-abdominal haemorrhage | Spinal subdural haemorrhage |
| Cerebellar haematoma | Intracerebral haematoma evacuation | Spleen contusion |

| Cerebellar haemorrhage | Intracranial haematoma | Splenic artery perforation |
|---|---|---|
| Cerebellar microhaemorrhage | Intracranial haemorrhage neonatal | Splenic haematoma |
| Cerebral aneurysm perforation | Intracranial tumour haemorrhage | Splenic haemorrhage |
| Cerebral aneurysm ruptured syphilitic | Intraocular haematoma | Splenic varices haemorrhage |
| Cerebral arteriovenous malformation haemorrhagic | Intrapartum haemorrhage | Splinter haemorrhages |
| Cerebral artery perforation | Intratumoural haematoma | Spontaneous haematoma |
| Cerebral cyst haemorrhage | Intraventricular haemorrhage | Spontaneous haemorrhage |
| Cerebral haematoma | Intraventricular haemorrhage neonatal | Stoma site haemorrhage |
| Cerebral haemorrhage | Iris haemorrhage | Stomatitis haemorrhagic |
| Cerebral haemorrhage foetal | Joint microhaemorrhage | Subarachnoid haematoma |
| Cerebral haemorrhage neonatal | Jugular vein haemorrhage | Subarachnoid haemorrhage |
| Cerebral microhaemorrhage | Kidney contusion | Subarachnoid haemorrhage neonatal |
| Cervix haematoma uterine | Lacrimal haemorrhage | Subcapsular hepatic haematoma |
| Cervix haemorrhage uterine | Large intestinal haemorrhage | Subcapsular renal haematoma |
| Chest wall haematoma | Large intestinal ulcer haemorrhage | Subcapsular splenic haematoma |
| Choroidal haematoma | Laryngeal haematoma | Subchorionic haematoma |
| Choroidal haemorrhage | Laryngeal haemorrhage | Subchorionic haemorrhage |
| Chronic gastrointestinal bleeding | Lip haematoma | Subclavian artery perforation |
| Chronic pigmented purpura | Lip haemorrhage | Subclavian vein perforation |
| Ciliary body haemorrhage | Liver contusion | Subcutaneous haematoma |
| Coital bleeding | Lower gastrointestinal haemorrhage | Subdural haematoma |
| Colonic haematoma | Lower limb artery perforation | Subdural haematoma evacuation |
| Conjunctival haemorrhage | Lymph node haemorrhage | Subdural haemorrhage |
| Contusion | Mallory-Weiss syndrome | Subdural haemorrhage neonatal |
| Corneal bleeding | Mediastinal haematoma | Subendocardial haemorrhage |
| Cullen's sign | Mediastinal haemorrhage | Subgaleal haematoma |
| Cystitis haemorrhagic | Medical device site bruise | Subgaleal haemorrhage |
| Deep dissecting haematoma | Medical device site haematoma | Subretinal haematoma |
| Diarrhoea haemorrhagic | Medical device site haemorrhage | Superior vena cava perforation |
| Disseminated intravascular coagulation | Melaena | Testicular haemorrhage |
| Diverticulitis intestinal haemorrhagic | Melaena neonatal | Thalamus haemorrhage |
| Diverticulum intestinal haemorrhagic | Meningorrhagia | Third stage postpartum haemorrhage |
| Duodenal ulcer haemorrhage | Menometrorrhagia | Thoracic haemorrhage |
| Duodenitis haemorrhagic | Mesenteric haematoma | Thrombocytopenic purpura |
| Ear haemorrhage | Mesenteric haemorrhage | Thrombomodulin increased |
| Ecchymosis | Mouth haemorrhage | Thrombotic thrombocytopenic purpura |
| Encephalitis haemorrhagic | Mucocutaneous haemorrhage | Thyroid haemorrhage |
| Enterocolitis haemorrhagic | Mucosal haemorrhage | Tongue haematoma |

| Epidural haemorrhage | Muscle contusion | Tongue haemorrhage |
|---|---|---|
| Epistaxis | Muscle haemorrhage | Tonsillar haemorrhage |
| Exsanguination | Myocardial haemorrhage | Tooth pulp haemorrhage |
| Extra-axial haemorrhage | Myocardial rupture | Tooth socket haemorrhage |
| Extradural haematoma | Naevus haemorrhage | Tracheal haemorrhage |
| Extradural haematoma evacuation | Nail bed bleeding | Traumatic haematoma |
| Extravasation blood | Nasal septum haematoma | Traumatic haemorrhage |
| Eye contusion | Neonatal gastrointestinal haemorrhage | Traumatic haemothorax |
| Eye haematoma | Nephritis haemorrhagic | Traumatic intracranial haematoma |
| Eye haemorrhage | Nipple exudate bloody | Traumatic intracranial haemorrhage |
| Eyelid bleeding | Occult blood positive | Tumour haemorrhage |
| Eyelid contusion | Ocular retrobulbar haemorrhage | Ulcer haemorrhage |
| Eyelid haematoma | Oesophageal haemorrhage | Umbilical cord haemorrhage |
| Femoral artery perforation | Oesophageal intramural haematoma | Umbilical haematoma |
| Femoral vein perforation | Oesophageal ulcer haemorrhage | Umbilical haemorrhage |
| Foetal-maternal haemorrhage | Oesophageal varices haemorrhage | Upper gastrointestinal haemorrhage |
| Fothergill sign positive | Oesophagitis haemorrhagic | Ureteric haemorrhage |
| Gallbladder haematoma | Omental haemorrhage | Urethral haemorrhage |
| Gastric haemorrhage | Optic disc haemorrhage | Urinary bladder haematoma |
| Gastric occult blood positive | Optic nerve sheath haemorrhage | Urinary bladder haemorrhage |
| Gastric ulcer haemorrhage | Oral blood blister | Urinary occult blood |
| Gastric ulcer haemorrhage, obstructive | Oral contusion | Urinary occult blood positive |
| Gastric varices haemorrhage | Oral mucosa haematoma | Urogenital haemorrhage |
| Gastritis alcoholic haemorrhagic | Oral purpura | Uterine haematoma |
| Gastritis haemorrhagic | Orbital haematoma | Uterine haemorrhage |
| Gastroduodenal haemorrhage | Orbital haemorrhage | Vaccination site bruising |
| Gastrointestinal anastomotic haemorrhage | Osteorrhagia | Vaccination site haematoma |
| Gastrointestinal haemorrhage | Ovarian haematoma | Vaccination site haemorrhage |
| Gastrointestinal polyp haemorrhage | Ovarian haemorrhage | Vaginal haematoma |
| Gastrointestinal ulcer haemorrhage | Palpable purpura | Vaginal haemorrhage |
| Gastrointestinal vascular malformation | | |
| haemorrhagic | Pancreatic haemorrhage | Varicose vein ruptured |
| Genital contusion | Pancreatic pseudocyst haemorrhage | Vascular access site bruising |
| Genital haemorrhage | Pancreatitis haemorrhagic | Vascular access site haematoma |
| Gingival bleeding | Papillary muscle haemorrhage | Vascular access site haemorrhage |
| Graft haemorrhage | Paranasal sinus haematoma | Vascular access site rupture |
| Grey Turner's sign | Paranasal sinus haemorrhage | Vascular anastomotic haemorrhage |
| Haemangioma rupture | Parathyroid haemorrhage | Vascular graft haemorrhage |

| Haemarthrosis | Parotid gland haemorrhage | Vascular pseudoaneurysm ruptured |
|---|---|---|
| Haematemesis | Pelvic haematoma | Vascular purpura |
| Haematochezia | Pelvic haematoma obstetric | Vascular rupture |
| Haematocoele | Pelvic haemorrhage | Vein rupture |
| Haematoma | Penile contusion | Venous haemorrhage |
| Haematoma evacuation | Penile haematoma | Venous perforation |
| Haematoma infection | Penile haemorrhage | Ventricle rupture |
| Haematoma muscle | Peptic ulcer haemorrhage | Vertebral artery perforation |
| Haematosalpinx | Pericardial haemorrhage | Vessel puncture site bruise |
| Haematospermia | Perineal haematoma | Vessel puncture site haematoma |
| Haematotympanum | Periorbital haematoma | Vessel puncture site haemorrhage |
| Haematuria | Periorbital haemorrhage | Vitreous haematoma |
| Haematuria traumatic | Periosteal haematoma | Vitreous haemorrhage |
| Haemobilia | Peripartum haemorrhage | Vulval haematoma |
| Haemoperitoneum | Peripheral artery aneurysm rupture | Vulval haematoma evacuation |
| Haemophilic arthropathy | Peripheral artery haematoma | Vulval haemorrhage |
| | Peripheral exudative haemorrhagic | |
| | chorioretinopathy | Withdrawal bleed |
| | • | Wound haematoma |
| | | Wound haemorrhage |
| | AESI Category: Gastrointestinal perforation | |
| Abdominal abscess | Enterocutaneous fistula | Mesenteric abscess |
| Abdominal hernia perforation | Enterovesical fistula | Neonatal intestinal perforation |
| Abdominal wall abscess | Fistula of small intestine | Oesophageal abscess |
| Abscess intestinal | Focal peritonitis | Oesophageal fistula |
| Acquired tracheo-oesophageal fistula | Gastric fistula | Pancreatic fistula repair |
| Anal abscess | Gastric fistula repair | Peptic ulcer perforation |
| Anal fistula | Gastric perforation | Peptic ulcer perforation, obstructive |
| Anal fistula infection | Gastric ulcer perforation | Peptic ulcer repair |
| Anal fistula repair | Gastric ulcer perforation, obstructive | Perforated ulcer |
| Anastomotic ulcer perforation | Gastrointestinal anastomotic leak | Perineal abscess |
| Anovulvar fistula | Gastrointestinal fistula | Perirectal abscess |
| Aorto-oesophageal fistula | Gastrointestinal fistula repair | Peritoneal abscess |
| Aortoenteric fistula | Gastrointestinal perforation | Peritoneocutaneous fistula |
| Appendiceal abscess | Gastrointestinal ulcer perforation | Peritonitis |
| Appendicitis perforated | Gastropleural fistula | Peritonitis bacterial |
| Arterioenteric fistula | Gastrosplenic fistula | Pneumoperitoneum |

| Atrio-oesophageal fistula | Ileal perforation | Pneumoretroperitoneum |
|---|---|---|
| Chemical peritonitis | Ileal ulcer perforation | Procedural intestinal perforation |
| Colo-urethral fistula | Incisional hernia perforation | Rectal abscess |
| Colon fistula repair | Inguinal hernia perforation | Rectal fistula repair |
| Colonic abscess | Intestinal fistula | Rectal perforation |
| Colonic fistula | Intestinal fistula infection | Rectoprostatic fistula |
| Diverticular fistula | Intestinal fistula repair | Rectourethral fistula |
| Diverticular perforation | Intestinal perforation | Retroperitoneal abscess |
| Diverticulitis intestinal perforated | Intestinal ulcer perforation | Small intestinal perforation |
| Douglas' abscess | Jejunal perforation | Small intestinal ulcer perforation |
| Duodenal perforation | Jejunal ulcer perforation | Spontaneous bacterial peritonitis |
| Duodenal rupture | Large intestinal ulcer perforation | Umbilical hernia perforation |
| Duodenal ulcer perforation | Large intestine perforation | Upper gastrointestinal perforation |
| Duodenal ulcer perforation, obstructive | Lower gastrointestinal perforation | |
| Duodenal ulcer repair | | |
| Enterocolonic fistula | | |
| | AESI Category: Embolic and thrombotic ev | |
| Acute aortic syndrome | Embolism venous | Prosthetic cardiac valve thrombosis |
| Acute coronary syndrome | Endarterectomy | Prosthetic vessel implantation |
| Acute myocardial infarction | Eye infarction | Pseudo-occlusion of internal carotid artery |
| Administration site thrombosis | Femoral artery embolism | Pulmonary artery occlusion |
| Adrenal thrombosis | Fluorescence angiogram abnormal | Pulmonary artery therapeutic procedure |
| Amaurosis | Foetal cerebrovascular disorder | Pulmonary artery thrombosis |
| Amaurosis fugax | Foetal vascular malperfusion | Pulmonary embolism |
| Aneurysm thrombosis | Gastric infarction | Pulmonary endarterectomy |
| Angiogram abnormal | Graft thrombosis | Pulmonary infarction |
| Angiogram cerebral abnormal | Haemorrhagic adrenal infarction | Pulmonary microemboli |
| Angiogram peripheral abnormal | Haemorrhagic cerebral infarction | Pulmonary thrombosis |
| Angioplasty | Haemorrhagic infarction | Pulmonary tumour thrombotic microangiopathy |
| Antiphospholipid syndrome | Haemorrhagic stroke | Pulmonary vein occlusion |
| Aortic bypass | Haemorrhagic transformation stroke | Pulmonary veno-occlusive disease |
| Aortic embolus | Haemorrhoids thrombosed | Pulmonary venous thrombosis |
| Aortic surgery | Hemiparesis | Quadriparesis |
| Aortic thrombosis | Hemiplegia | Quadriplegia |
| Aortogram abnormal | Heparin-induced thrombocytopenia | Renal artery angioplasty |
| Application site thrombosis | Hepatic artery embolism | Renal artery occlusion |
| Arterectomy | Hepatic artery occlusion | Renal artery thrombosis |

| Arterectomy with graft replacement | Hepatic artery thrombosis | Renal embolism |
|---|---|---|
| Arterial angioplasty | Hepatic infarction | Renal infarct |
| Arterial bypass operation | Hepatic vascular thrombosis | Renal vascular thrombosis |
| Arterial graft | Hepatic vein embolism | Renal vein embolism |
| Arterial occlusive disease | Hepatic vein occlusion | Renal vein occlusion |
| Arterial revascularisation | Hepatic vein thrombosis | Renal vein thrombosis |
| Arterial stent insertion | Homans' sign positive | Renal-limited thrombotic microangiopathy |
| Arterial therapeutic procedure | Hypothenar hammer syndrome | Retinal artery embolism |
| Arterial thrombosis | Iliac artery embolism | Retinal artery occlusion |
| Arteriogram abnormal | Iliac artery occlusion | Retinal artery thrombosis |
| Arteriogram carotid abnormal | Iliac vein occlusion | Retinal infarction |
| Arteriotomy | Implant site thrombosis | Retinal vascular thrombosis |
| Arteriovenous fistula occlusion | Incision site vessel occlusion | Retinal vein occlusion |
| Arteriovenous fistula thrombosis | Infarction | Retinal vein thrombosis |
| Arteriovenous graft thrombosis | Inferior vena cava syndrome | Revascularisation procedure |
| Artificial blood vessel occlusion | Inferior vena caval occlusion | SI QIII TIII pattern |
| Aseptic cavernous sinus thrombosis | Infusion site thrombosis | Segmental arterial mediolysis |
| Atherectomy | Injection site thrombosis | Shunt occlusion |
| Atherosclerotic plaque rupture | Inner ear infarction | Shunt thrombosis |
| Atrial appendage closure | Instillation site thrombosis | Sigmoid sinus thrombosis |
| Atrial appendage resection | Internal capsule infarction | Silent myocardial infarction |
| Atrial thrombosis | Intestinal infarction | Spinal artery embolism |
| Autoimmune heparin-induced thrombocytopenia | Intra-aortic balloon placement | Spinal artery thrombosis |
| Axillary vein thrombosis | Intracardiac mass | Spinal cord infarction |
| Basal ganglia infarction | Intracardiac thrombus | Spinal stroke |
| Basal ganglia stroke | Intraoperative cerebral artery occlusion | Splenic artery thrombosis |
| Basilar artery occlusion | Ischaemic cerebral infarction | Splenic embolism |
| Basilar artery thrombosis | Ischaemic stroke | Splenic infarction |
| Blindness transient | Jugular vein embolism | Splenic thrombosis |
| Bone infarction | Jugular vein occlusion | Splenic vein occlusion |
| Brachiocephalic artery occlusion | Jugular vein thrombosis | Splenic vein thrombosis |
| | | Spontaneous heparin-induced thrombocytopenia |
| Brachiocephalic vein occlusion | Lacunar infarction | syndrome |
| Brachiocephalic vein thrombosis | Lambl's excrescences | Stoma site thrombosis |
| Brain stem embolism | Left atrial appendage closure implant | Stress cardiomyopathy |
| Brain stem infarction | Leriche syndrome | Stroke in evolution |
| Brain stem stroke | Mahler sign | Strokectomy |
| Brain stem thrombosis | May-Thurner syndrome | Subclavian artery embolism |

| Budd-Chiari syndrome | Medical device site thrombosis | Subclavian artery occlusion |
|---|---|---|
| Capsular warning syndrome | Mesenteric arterial occlusion | Subclavian artery thrombosis |
| Cardiac ventricular thrombosis | Mesenteric arteriosclerosis | Subclavian vein occlusion |
| Carotid angioplasty | Mesenteric artery embolism | Subclavian vein thrombosis |
| Carotid arterial embolus | Mesenteric artery stenosis | Superficial vein thrombosis |
| Carotid artery bypass | Mesenteric artery stent insertion | Superior sagittal sinus thrombosis |
| Carotid artery occlusion | Mesenteric artery thrombosis | Superior vena cava occlusion |
| Carotid artery stent insertion | Mesenteric vascular insufficiency | Superior vena cava syndrome |
| Carotid artery thrombosis | Mesenteric vascular occlusion | Surgical vascular shunt |
| Carotid endarterectomy | Mesenteric vein thrombosis | Testicular infarction |
| Catheter directed thrombolysis | Mesenteric venous occlusion | Thalamic infarction |
| Catheter site thrombosis | Metabolic stroke | Thrombectomy |
| Catheterisation venous | Microembolism | Thromboangiitis obliterans |
| Cavernous sinus thrombosis | Monoparesis | Thromboembolectomy |
| Central venous catheterisation | Monoplegia | Thrombolysis |
| Cerebellar artery occlusion | Muscle infarction | Thrombophlebitis |
| Cerebellar artery thrombosis | Myocardial infarction | Thrombophlebitis migrans |
| Cerebellar embolism | Myocardial necrosis | Thrombophlebitis neonatal |
| Cerebellar infarction | Obstetrical pulmonary embolism | Thrombosed varicose vein |
| Cerebral artery embolism | Obstructive shock | Thrombosis |
| Cerebral artery occlusion | Ophthalmic artery occlusion | Thrombosis corpora cavernosa |
| Cerebral artery stent insertion | Ophthalmic artery thrombosis | Thrombosis in device |
| Cerebral artery thrombosis | Ophthalmic vein thrombosis | Thrombosis mesenteric vessel |
| Cerebral congestion | Optic nerve infarction | Thrombosis prophylaxis |
| Cerebral hypoperfusion | Ovarian vein thrombosis | Thrombosis with thrombocytopenia syndrome |
| Cerebral infarction | Paget-Schroetter syndrome | Thrombotic cerebral infarction |
| Cerebral infarction foetal | Pancreatic infarction | Thrombotic microangiopathy |
| Cerebral ischaemia | Papillary muscle infarction | Thrombotic stroke |
| Cerebral microembolism | Paradoxical embolism | Thrombotic thrombocytopenic purpura |
| Cerebral microinfarction | Paraneoplastic thrombosis | Thyroid infarction |
| Cerebral septic infarct | Paraparesis | Transient ischaemic attack |
| Cerebral thrombosis | Paraplegia | Transverse sinus thrombosis |
| Cerebral vascular occlusion | Paresis | Truncus coeliacus thrombosis |
| Cerebral venous sinus thrombosis | Pelvic venous thrombosis | Tumour embolism |
| Cerebral venous thrombosis | Penile artery occlusion | Tumour thrombectomy |
| Cerebrospinal thrombotic tamponade | Penile vein thrombosis | Tumour thrombosis |
| Cerebrovascular accident | Percutaneous coronary intervention | Ultrasonic angiogram abnormal |
| Cerebrovascular accident prophylaxis | Peripheral arterial occlusive disease | Ultrasound Doppler abnormal |

| Cerebrovascular disorder | Peripheral arterial reocclusion | Umbilical cord occlusion |
|---|---|---|
| Cerebrovascular insufficiency | Peripheral artery angioplasty | Umbilical cord thrombosis |
| Cerebrovascular operation | Peripheral artery bypass | Vaccination site thrombosis |
| Cerebrovascular stenosis | Peripheral artery occlusion | Vascular access site thrombosis |
| Choroidal infarction | Peripheral artery stent insertion | Vascular device occlusion |
| Coeliac artery occlusion | Peripheral artery surgery | Vascular graft |
| Collateral circulation | Peripheral artery thrombosis | Vascular graft occlusion |
| Compression garment application | Peripheral embolism | Vascular graft thrombosis |
| Coronary angioplasty | Peripheral endarterectomy | Vascular operation |
| Coronary arterial stent insertion | Peripheral revascularisation | Vascular pseudoaneurysm thrombosis |
| Coronary artery bypass | Peripheral vein occlusion | Vascular stent insertion |
| Coronary artery embolism | Peripheral vein thrombosis | Vascular stent occlusion |
| Coronary artery occlusion | Peripheral vein thrombus extension | Vascular stent thrombosis |
| Coronary artery reocclusion | Phlebectomy | Vasodilation procedure |
| Coronary artery surgery | Pituitary infarction | Vena cava embolism |
| Coronary artery thrombosis | Placental infarction | Vena cava filter insertion |
| Coronary bypass thrombosis | Pneumatic compression therapy | Vena cava filter removal |
| Coronary endarterectomy | Popliteal artery entrapment syndrome | Vena cava thrombosis |
| Coronary revascularisation | Portal shunt procedure | Venogram abnormal |
| Coronary vascular graft occlusion | Portal vein cavernous transformation | Venoocclusive disease |
| Deep vein thrombosis | Portal vein embolism | Venoocclusive liver disease |
| Deep vein thrombosis postoperative | Portal vein occlusion | Venous angioplasty |
| Device embolisation | Portal vein thrombosis | Venous occlusion |
| Device occlusion | Portosplenomesenteric venous thrombosis | Venous operation |
| Device related thrombosis | Post procedural myocardial infarction | Venous recanalisation |
| Diplegia | Post procedural pulmonary embolism | Venous repair |
| Directional Doppler flow tests abnormal | Post procedural stroke | Venous stent insertion |
| Disseminated intravascular coagulation | Post thrombotic syndrome | Venous thrombosis |
| Disseminated intravascular coagulation in newborn | Postinfarction angina | Venous thrombosis in pregnancy |
| Embolia cutis medicamentosa | Postoperative thrombosis | Venous thrombosis limb |
| Embolic cerebellar infarction | Postpartum thrombosis | Venous thrombosis neonatal |
| Embolic cerebral infarction | Postpartum venous thrombosis | Vertebral artery occlusion |
| Embolic pneumonia | Precerebral artery embolism | Vertebral artery thrombosis |
| Embolic stroke | Precerebral artery occlusion | Vessel puncture site occlusion |
| Embolism | Precerebral artery thrombosis | Vessel puncture site thrombosis |
| Embolism arterial | Profundaplasty | Visceral venous thrombosis |
| | • ′ | Visual acuity reduced transiently |
| | | Visual midline shift syndrome |

| | AESI Category: Hepatic function abnormal | |
|---|---|---|
| AST/ALT ratio abnormal | Gastric variceal injection | Hypofibrinogenaemia |
| Acquired antithrombin III deficiency | Gastric variceal ligation | Hypoprothrombinaemia |
| Acquired factor IX deficiency | Gastric varices | Hypothrombinaemia |
| Acquired factor V deficiency | Gastric varices haemorrhage | Hypothromboplastinaemia |
| | Gastrooesophageal variceal haemorrhage | |
| Acquired factor VIII deficiency | prophylaxis | Icterus index increased |
| Acquired factor XI deficiency | Graft versus host disease in liver | Immune-mediated cholangitis |
| Acquired hepatocerebral degeneration | Guanase increased | Immune-mediated hepatic disorder |
| Acquired protein S deficiency | Haemangioma of liver | Immune-mediated hepatitis |
| Acute graft versus host disease in liver | Haemorrhagic hepatic cyst | International normalised ratio abnormal |
| Acute hepatic failure | Hepaplastin abnormal | International normalised ratio increased |
| Acute on chronic liver failure | Hepaplastin decreased | Intestinal varices |
| Acute yellow liver atrophy | Hepatectomy | Intestinal varices haemorrhage |
| Alanine aminotransferase abnormal | Hepatic adenoma | Ischaemic hepatitis |
| Alanine aminotransferase increased | Hepatic angiosarcoma | Jaundice |
| Allergic hepatitis | Hepatic artery flow decreased | Jaundice cholestatic |
| Alloimmune hepatitis | Hepatic atrophy | Jaundice hepatocellular |
| Ammonia abnormal | Hepatic calcification | Kayser-Fleischer ring |
| Ammonia increased | Hepatic cancer | Liver carcinoma ruptured |
| Anti factor X activity abnormal | Hepatic cancer metastatic | Liver dialysis |
| Anti factor X activity decreased | Hepatic cancer recurrent | Liver disorder |
| Anti factor X activity increased | Hepatic cancer stage I | Liver function test abnormal |
| Anti-liver cytosol antibody type 1 positive | Hepatic cancer stage II | Liver function test decreased |
| Antithrombin III decreased | Hepatic cancer stage III | Liver function test increased |
| Ascites | Hepatic cancer stage IV | Liver induration |
| Aspartate aminotransferase abnormal | Hepatic cirrhosis | Liver injury |
| Aspartate aminotransferase increased | Hepatic cyst | Liver operation |
| Asterixis | Hepatic cyst ruptured | Liver palpable |
| Autoimmune hepatitis | Hepatic cytolysis | Liver scan abnormal |
| Bacterascites | Hepatic encephalopathy | Liver tenderness |
| Benign hepatic neoplasm | Hepatic encephalopathy prophylaxis | Liver transplant |
| Benign hepatobiliary neoplasm | Hepatic enzyme abnormal | Liver-kidney microsomal antibody positive |
| Bile output abnormal | Hepatic enzyme decreased | Lupoid hepatic cirrhosis |
| Bile output decreased | Hepatic enzyme increased | Lupus hepatitis |
| • | | Magnetic resonance imaging hepatobiliary |
| Biliary ascites | Hepatic failure | abnormal |

| | | Magnetic resonance proton density fat fraction |
|---|---|---|
| Biliary cirrhosis | Hepatic fibrosis | measurement |
| | | Mitochondrial aspartate aminotransferase |
| Biliary fibrosis | Hepatic function abnormal | increased |
| Bilirubin conjugated abnormal | Hepatic haemangioma rupture | Mixed hepatocellular cholangiocarcinoma |
| Bilirubin conjugated increased | Hepatic hamartoma | Mixed liver injury |
| | | Molar ratio of total branched-chain amino acid |
| Bilirubin excretion disorder | Hepatic hydrothorax | to tyrosine |
| Bilirubin urine present | Hepatic hypertrophy | Nodular regenerative hyperplasia |
| Biopsy liver abnormal | Hepatic hypoperfusion | Non-alcoholic fatty liver |
| Blood bilirubin abnormal | Hepatic infiltration eosinophilic | Non-alcoholic steatohepatitis |
| Blood bilirubin increased | Hepatic lesion | Non-cirrhotic portal hypertension |
| Blood bilirubin unconjugated increased | Hepatic lipoma | Ocular icterus |
| Blood fibrinogen abnormal | Hepatic mass | Oedema due to hepatic disease |
| Blood fibrinogen decreased | Hepatic necrosis | Oesophageal varices haemorrhage |
| Blood thrombin abnormal | Hepatic neoplasm | Omental oedema |
| Blood thrombin decreased | Hepatic neuroendocrine tumour | Parenteral nutrition associated liver disease |
| Blood thromboplastin abnormal | Hepatic pain | Perihepatic discomfort |
| Blood thromboplastin decreased | Hepatic sarcoma | Peripancreatic varices |
| Bromosulphthalein test abnormal | Hepatic sequestration | Portal fibrosis |
| Cardiohepatic syndrome | Hepatic steato-fibrosis | Portal hypertension |
| Child-Pugh-Turcotte score abnormal | Hepatic steatosis | Portal hypertensive colopathy |
| Child-Pugh-Turcotte score increased | Hepatic vascular resistance increased | Portal hypertensive enteropathy |
| Cholaemia | Hepatic venous pressure gradient abnormal | Portal hypertensive gastropathy |
| Cholangiosarcoma | Hepatic venous pressure gradient increased | Portal vein cavernous transformation |
| Cholestasis | Hepatitis | Portal vein dilatation |
| Cholestatic liver injury | Hepatitis acute | Portopulmonary hypertension |
| Cholestatic pruritus | Hepatitis cholestatic | Primary biliary cholangitis |
| Chronic graft versus host disease in liver | Hepatitis chronic active | Protein C decreased |
| Chronic hepatic failure | Hepatitis chronic persistent | Protein S abnormal |
| Chronic hepatitis | Hepatitis fulminant | Protein S decreased |
| Coagulation factor IX level abnormal | Hepatitis toxic | Prothrombin level abnormal |
| Coagulation factor IX level decreased | Hepatobiliary cancer | Prothrombin level decreased |
| Coagulation factor V level abnormal | Hepatobiliary cancer in situ | Prothrombin time abnormal |
| Coagulation factor V level decreased | Hepatobiliary cyst | Prothrombin time prolonged |
| Coagulation factor VII level abnormal | Hepatobiliary disease | Prothrombin time ratio abnormal |
| Coagulation factor VII level decreased | Hepatobiliary neoplasm | Prothrombin time ratio increased |
| Coagulation factor X level abnormal | Hepatobiliary scan abnormal | Radiation hepatitis |

| Coagulation factor X level decreased | Hepatoblastoma | Regenerative siderotic hepatic nodule |
|---|---|---|
| Coagulation factor decreased | Hepatoblastoma recurrent | Renal and liver transplant |
| Coma hepatic | Hepatocellular carcinoma | Retrograde portal vein flow |
| Computerised tomogram liver abnormal | Hepatocellular foamy cell syndrome | Reye's syndrome |
| Congestive hepatopathy | Hepatocellular injury | Reynold's syndrome |
| Cryptogenic cirrhosis | Hepatomegaly | Splenic varices |
| Diabetic hepatopathy | Hepatopulmonary syndrome | Splenic varices haemorrhage |
| Drug-induced liver injury | Hepatorenal failure | Spontaneous bacterial peritonitis |
| Duodenal varices | Hepatorenal syndrome | Steatohepatitis |
| Flood syndrome | Hepatosplenomegaly | Subacute hepatic failure |
| Focal nodular hyperplasia | Hepatotoxicity | Sugiura procedure |
| Foetor hepaticus | Hyperammonaemia | Thrombin time abnormal |
| Galactose elimination capacity test abnormal | Hyperbilirubinaemia | Thrombin time prolonged |
| Galactose elimination capacity test decreased | Hypercholia | Total bile acids increased |
| Gallbladder varices | Hyperfibrinolysis | Transaminases abnormal |
| Gamma-glutamyltransferase abnormal | Hypertransaminasaemia | Transaminases increased |
| Gamma-glutamyltransferase increased | Hypocoagulable state | Ultrasound liver abnormal |
| | | Urine bilirubin increased |
| | | Varices oesophageal |
| | | Varicose veins of abdominal wall |
| | | White nipple sign |
| | | X-ray hepatobiliary abnormal |
| | SI Category: Left ventricular ejection fractio | |
| Acute left ventricular failure | Cardiohepatic syndrome | Hepatojugular reflux |
| Acute pulmonary oedema | Cardiopulmonary failure | Left ventricular failure |
| Acute right ventricular failure | Cardiorenal syndrome | Low cardiac output syndrome |
| Cardiac asthma | Chronic left ventricular failure | Neonatal cardiac failure |
| Cardiac failure | Chronic right ventricular failure | Obstructive shock |
| Cardiac failure acute | Congestive hepatopathy | Pulmonary oedema |
| Cardiac failure chronic | Cor pulmonale | Pulmonary oedema neonatal |
| Cardiac failure congestive | Cor pulmonale acute | Radiation associated cardiac failure |
| Cardiac failure high output | Cor pulmonale chronic | Right ventricular ejection fraction decreased |
| Cardiogenic shock | Ejection fraction decreased | Right ventricular failure |
| | | Ventricular failure |

## Appendix 4: imAE by Preferred Term

| imAE Category: Immune-mediated AEs | | |
|---|---|---|
| Immune-mediated adrenal insufficiency | Immune-mediated endocrinopathy | Immune-mediated myositis |
| Immune-mediated adverse reaction | Immune-mediated enterocolitis | Immune-mediated nephritis |
| Immune-mediated arthritis | Immune-mediated gastritis | Immune-mediated neurological disorder |
| Immune-mediated cholangitis | Immune-mediated hepatic disorder | Immune-mediated neuropathy |
| Immune-mediated cholestasis | Immune-mediated hepatitis | Immune-mediated oesophagitis |
| Immune-mediated cystitis | Immune-mediated hyperthyroidism | Immune-mediated pancreatitis |
| Immune-mediated cytopenia | Immune-mediated hypophysitis | Immune-mediated renal disorder |
| Immune-mediated dermatitis | Immune-mediated hypothyroidism | Immune-mediated thyroiditis |
| Immune-mediated encephalitis | Immune-mediated lung disease | Immune-mediated uveitis |
| Immune-mediated encephalopathy | Immune-mediated myocarditis | |
| • • | imAE Category: Skin Adverse Reactio | ns |
| Acute febrile neutrophilic dermatosis | Oculomucocutaneous syndrome | Urticaria papular |
| Angioedema | Pruritus | Urticaria vesiculosa |
| Blister | Rash | Vitiligo |
| Cutaneous vasculitis | Rash erythematous | Acute generalised exanthematous pustulosis |
| Dermatitis | Rash follicular | Urticarial vasculitis |
| Dermatitis allergic | Rash macular | Rash maculovesicular |
| Dermatitis bullous | Rash maculo-papular | Urticaria chronic |
| Dermatitis exfoliative | Rash papular | Mucocutaneous rash |
| Dermatitis exfoliative generalised | Rash pruritic | Toxic skin eruption |
| Drug eruption | Rash pustular | Dermatitis psoriasiform |
| Eczema | Rash vesicular | Epidermal necrosis |
| Erythema multiforme | Skin depigmentation | Mucosal exfoliation |
| Fixed eruption | Skin exfoliation | Exfoliative rash |
| Idiopathic urticaria | Skin hypopigmentation | Mucosal necrosis |
| Leukoderma | Skin necrosis | Drug reaction with eosinophilia and systemic symptoms |
| Mucocutaneous ulceration | Stevens-Johnson syndrome | Autoimmune dermatitis |
| Mucosal ulceration | Toxic epidermal necrolysis | Nodular rash |
| Oculomucocutaneous syndrome | Urticaria | |
| imAE Category: Diabetes | | |
| Diabetes mellitus | Diabetic ketoacidosis | Ketosis-prone diabetes mellitus |
| Diabetes mellitus inadequate control | Diabetic ketoacidotic hyperglycaemic coma | Pancreatogenous diabetes |
| Diabetes with hyperosmolarity | Diabetic ketosis | Latent autoimmune diabetes in adults |
| Diabetic hyperglycaemic coma | Increased insulin requirement | Type 1 diabetes mellitus |
| Diabetic hyperosmolar coma | Insulin resistant diabetes | Fulminant type 1 diabetes mellitus |

Appendix 5: MedDRA (Version 25.0) Preferred Term List for COVID-19 Related AE

| Asymptomatic COVID-19 | Occupational exposure to SARS-CoV-2 |
|---|---|
| Breakthrough COVID-19 | Post-acute COVID-19 syndrome |
| Congenital COVID-19 | SARS-CoV-2 antibody test positive |
| Coronavirus infection | SARS-CoV-2 carrier |
| Coronavirus pneumonia | SARS-CoV-2 RNA decreased |
| Coronavirus test positive | SARS-CoV-2 RNA fluctuation |
| COVID-19 | SARS-CoV-2 RNA increased |
| COVID-19 immunisation | SARS-CoV-2 sepsis |
| COVID-19 pneumonia | SARS-CoV-2 test false negative |
| COVID-19 prophylaxis | SARS-CoV-2 test positive |
| COVID-19 treatment | SARS-CoV-2 viraemia |
| Exposure to SARS-CoV-2 | Suspected COVID-19 |
| Multisystem inflammatory syndrome | Thrombosis with thrombocytopenia syndrome |
| Multisystem inflammatory syndrome in adults | Vaccine derived SARS-CoV-2 infection |
| Multisystem inflammatory syndrome in children | |

## Appendix 6 : Conversion tables for urinalysis results

| Blood/Leucocytes (for parameter red blood cell and white blood cell) | | |
|---|---|---|
| Negative | 0 | 0 cells/μL |
| Trace | 1+ | 1-24 cells/μL |
| Small | 2+ | 25-79 cells/μL |
| Medium | 3+ | 80-199 cells/μL |
| Large | 4+ | ≥ 200 cells/μL |

| Proteinuria (for parameter protein) | | | | |
|---|---|---|---|---|
| NCI-CTCAE | Protein by urinalysis | 24-hour protein quantitation | Protein by urinalysis | 24-hour protein quantitation |
| Grade | | | | |
| 0 | 0 | | Negative | <10 mg/dL |
| 1 | 1+ | <1.0g | Trace | 11 <b>-</b> 99 mg/dL |
| 2 | 2+ | <2.0g | Small | 99-299 mg/dL |
| 2 | ≥2+ | <3.5 g (excluding 3.5 g) | Medium | 300-999 mg/dL |
| 3 | 4+ | ≥3.5 g | large | >1000 mg/dL |

# hmp-2020-013-00us3-7015654-statistical analysis plan v2.0 Final 29Jul2024

Final Audit Report 2024-07-31

| Created: | 2024-07-29 |
|-----------------|------------|
| Ву: | PPD |
| Status: | Signed |
| Transaction ID: | PPD |

# "hmp-2020-013-00us3-7015654-statistical analysis plan v2.0 Fin al 29Jul2024" History

| 1 | Document created by PPD | |
|---|---|---|
| | 2024-07-29 - 9:57:59 PM GMT- IP address: PPD | |
| <b>②</b> | PPD authenticated with Adobe Acrobat S | Sign. |
| | Challenge: The user completed the signing ceremony. | |
| | 2024-07-29 - 10:03:41 PM GMT | |
| do | Document e-signed by PPD | |
| | Signing reason: I am the author | |
| | Signature Date: 2024-07-29 - 10:03:43 PM GMT - Time Source: server- IP address: PPD | |
| | Document emailed to PPD | |
| | PPD for signature | |
| | 2024-07-29 - 10:03:45 PM GMT | |
| 3 | Email viewed by PPD | |
| | 2024-07-30 - 1:53:41 PM GMT- IP address PPD | |
| 0 | PPD | authenticate |
| | with Adobe Acrobat Sign. | |
| | Challenge: The user completed the signing ceremony. | |
| | 2024-07-30 - 1:56:09 PM GMT | |
| do | Document e-signed by PPD | |
| | PPD | |
| | Signing reason: I am the approver | |
| | Signature Date: 2024-07-30 - 1:56:11 PM GMT - Time Source: server- IP address: PPD | |



Document emailed to PPD PPD for signature

2024-07-30 - 1:56:13 PM GMT

Email viewed by PPD

2024-07-31 - 3:11:41 AM GMT- IP address PPD

PPD authenticated

with Adobe Acrobat Sign.

Challenge: The user completed the signing ceremony.

2024-07-31 - 3:14:11 AM GMT

Document e-signed by PPD PPD

Signing reason: I am the approver

Signature Date: 2024-07-31 - 3:14:14 AM GMT - Time Source: server- IP address: PPD

Agreement completed.
 2024-07-31 - 3:14:14 AM GMT



# hmp-2020-013-00us3-7015654-statistical analysis plan v2.0 Final 29Jul2024

Final Audit Report 2024-07-31

| Status: Signed | Created: | 2024-07-31<br>PPD |
|----------------|-------------------------|-------------------|
| DDD | Ву: | |
| | Status: Transaction ID: | Signed PPD |

# "hmp-2020-013-00us3-7015654-statistical analysis plan v2.0 Fin al 29Jul2024" History

| 60 | Document digitally presigned by Adobe Acre<br>2024-07-31 - 6:55:50 AM GMT- IP address: PPD | robat Sign (acrobat-sign-certified@adobe.com) |
|---|---|---|
| 1 | Document created by PPD 2024-07-31 - 11:33:57 AM GMT- IP address: PPD | |
| do | Signer PPD 2024-07-31 - 11:35:12 AM GMT- IP address: PPD | entered name at signing as PPD |
| 0 | PPD Challenge: The user completed the signing ceremony. 2024-07-31 - 11:35:13 AM GMT | authenticated with Adobe Acrobat Sign. |
| Ó | Document e-signed by PPD Signing reason: Approved Signature Date: 2024-07-31 - 11:35:14 AM GMT - Time | ne Source: server- IP address: PPD |
| E, | Document emailed to PPD 2024-07-31 - 11:35:16 AM GMT | for signature |
| 1 | Email viewed by PPD<br>2024-07-31 - 12:00:25 PM GMT- IP address: PPD | |
| 0 | Challenge: The user opened the agreement. | nticated with Adobe Acrobat Sign. |



PPD authenticated with Adobe Acrobat Sign. Challenge: The user completed the signing ceremony. 2024-07-31 - 12:01:37 PM GMT Document e-signed by PPD Signing reason: Approved Signature Date: 2024-07-31 - 12:01:38 PM GMT - Time Source: server- IP address: PPD Document emailed to PPD for signature 2024-07-31 - 12:01:41 PM GMT Email viewed by PPD 2024-07-31 - 12:03:09 PM GMT- IP address: PPD PPD authenticated with Adobe Acrobat Sign. Challenge: The user opened the agreement. 2024-07-31 - 12:03:39 PM GMT Document e-signed by PPD Signing reason: Approved Signature Date: 2024-07-31 - 12:04:14 PM GMT - Time Source: server- IP address: PPD

Agreement completed.

2024-07-31 - 12:04:14 PM GMT

PPD authenticated with Adobe Acrobat Sign.

Challenge: The user completed the signing ceremony.

2024-07-31 - 12:04:14 PM GMT

